CLINICAL TRIAL: NCT00153101
Title: ONTARGET ONgoing Telmisartan Alone and in Combination With Ramipril Global Endpoint Trial A Large, Simple Randomized Trial of an Angiotensin II Receptor Antagonist (Telmisartan) and an ACE-Inhibitor (Ramipril) in Patients at High Risk for Cardiovascular Events and TRANSCEND Telmisartan Randomized AssessmeNt Study in aCE iNtolerant Subjects With Cardiovascular Disease. A Parallel Study Comparing the Effects of Telmisartan With Placebo and Outcomes in Patients at High Risk for Cardiovascular Events and Intolerant to ACE-I.
Brief Title: Effectiveness and Safety of Ramipril Alone Compared With Telmisartan Alone and in Combination With Ramipril in Patients at High Risk for Cardiovascular Events. Patients Intolerant to Ramipril Were Entered in TRANSCEND, Telmisartan Compared to Placebo.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Prevention
Other Study IDs: 502.373; NCT00034931 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Telmisartan; Ramipril

INTERVENTIONS:
Drug: Telmisartan
Drug: Combination of Telmisartan and Ramipril
Drug: Ramipril

SUMMARY:
The Ongoing Telmisartan Alone and in combination wiht Ramipril Global Endpoint trial (ONTARGET): The primary objectives are to determine if (a) telmisartan 80mg daily and ramipril 10mg daily combination therapy is more effective in reducing the composite endpoint of Cardiovascular Death (CV) death, Myocardial infarction (MI), stroke or hospitalization for Congestive Heart Failure (CHF) compared with ramipril 10mg alone; and (b) telmisartan 80mg daily is at least as effective as (i.e. not less effective than) ramipril 10mg daily, on this endpoint.

Telmisartan Randomised Assessment Study in Angiotension converting Enzyme inhibitor intolerant subjects with Cardiovascular Disease. (TRANSCEND): The primary objective of the study is to determine if treatment with telmisartan 80mg daily is superior to placebo reducing the composite endpoint of Cardiovascular Death (CV), Myocardial Infarction ( MI)I, stroke or hospitalization for Congestive Heart Failure (CHF) in patients who are intolerant to Angiotension Converting Enzyme inhibitors.

ELIGIBILITY:
Inclusion Criteria:

Coronary Artery Disease: Previous Myocardial infarction(> 2 days prior to informed consent), or stable or previous unstable angina (> 30 days prior to informed consent) with documented multivessel coronary artery disease or a positive stress test, or multivessel Percutaneous Transluminal Coronary Angioplasty (> 30 days prior to informed consent), or previous multivessel Coronary Artery Bypass Grafting without angina (if surgery performed > 4 years prior to informed consent) or with recurrent angina after surgery.

Other High Risk:

1. Peripheral Arterial Disease: Previous limb bypass surgery or angioplasty or amputation, intermittent claudication on history with ankle/arm Blood Pressure ratio < 0.8 on at least one side, or significant stenosis by angiography or non-invasive testing
2. Previous stroke
3. Transient ischemic Attack > 7 days and < 1 year prior to informed consent
4. Diabetes Mellitus (types I or II): with evidence of end-organ damage (retinopathy, Left ventricular hypertrophy, micro or macro albuminuria), or any evidence of previous cardiac or vascular disease.

No definite and specific indication or contraindication for any of the study treatments. Written informed consent.

Exclusion Criteria:

A. Medication use:

1. Inability to discontinue Angiotension Converting Enzyme (ACE) inhibitors or Angiotension 2 receptor antagonists (AIIAs).
2. Patients with known hypersensitivity or intolerance to Angiotension 2 receptor antagonists (AIIAs) or Angiotension Converting Enzyme (ACE)inhibitors.

NOTE: Patients with known intolerance to Angiotension Converting Enzyme inhibitor intolerance ( ACE-I) can be enrolled in the TRANSCEND study.

B. Cardiovascular disease:

1. Symptomatic congestive heart failure.
2. Hemodynamically significant primary valvular or outflow tract obstruction (e.g. aortic or mitral valve stenosis, asymmetric septal hypertrophy, malfunctioning prosthetic valve).
3. Constrictive pericarditis.
4. Complex congenital heart disease.
5. Syncopal episodes of unknown etiology < 3 months before informed consent.
6. Planned cardiac surgery or angioplasty within three months.
7. Uncontrolled hypertension on treatment (i.e.Blood pressure ( BP) > 160/100).
8. Heart transplant recipient.
9. Strokes due to subarachnoid hemorrhage

C. Other conditions:

1. Significant renal disease defined as:

   1. Renal artery stenosis;
   2. Creatinine clearance < 0.6 ml/min or serum creatinine > 265 umol/L (> 3.0 mg/dL);
   3. Hyperkalemia: potassium > 5.5 mmol/L.
   4. Proteinuria* (for TRANSCEND only).
2. Hepatic dysfunction as defined by the following laboratory parameters: Serum Glutamate Pyruvate Transaminase( SGPT) Alaninaminotransferase (ALT) or Serum Glutamic Oxaloacetic Transaminase (SGOT) Aspartate aminotransferase (AST) > than 4 times upper limit of normal or additional criteria for hepatic impairment the upper limit of normal range, total Bilirubin > 20 umol/L, biliary obstructive disorders.
3. Uncorrected volume depletion or sodium depletion.
4. Primary aldosteronism.
5. Hereditary fructose intolerance.
6. Any other major non-cardiac illness expected to reduce life expectancy or interfere with study participation.
7. Patient is simultaneously taking another experimental drug.
8. Patient with significant disability that precludes regular attendance at clinic for follow-up.
9. Patient has sufficient disability or other incapacity that precludes regular attendance at clinic for follow-up.
10. Unable or unwilling to provide written informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31546 (Actual)
Dates: Start 2001-11; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (732):
- United States (100):
  - 502.373.0256 Boehringer Ingelheim Investigational Site, Athens, Alabama
  - 502.373.0251 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 502.373.0182 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 502.373.0188 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 502.373.0189 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 502.373.0177 Boehringer Ingelheim Investigational Site, Tuscon, Arizona
  - 502.373.0209 Boehringer Ingelheim Investigational Site, Bentonville, Arkansas
  - 502.373.0173 Boehringer Ingelheim Investigational Site, Concord, California
  - 502.373.0266 Boehringer Ingelheim Investigational Site, Harbor City, California
  - 502.373.0283 Boehringer Ingelheim Investigational Site, Loma Linda, California
  - 502.373.0180 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 502.373.0175 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 502.373.0165 Boehringer Ingelheim Investigational Site, San Diego, California
  - 502.373.0228 Boehringer Ingelheim Investigational Site, San Leandro, California
  - 502.373.0205 Boehringer Ingelheim Investigational Site, Sylmar, California
  - 502.373.0277 Boehringer Ingelheim Investigational Site, West Hills, California
  - 502.373.0226 Boehringer Ingelheim Investigational Site, Bridgeport, Connecticut
  - 502.373.0174 Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - 502.373.0258 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 502.373.0179 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 502.373.0183 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 502.373.0240 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 502.373.0171 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 502.373.0282 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 502.373.0214 Boehringer Ingelheim Investigational Site, Weston, Florida
  - 502.373.0161 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 502.373.0193 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 502.373.0201 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 502.373.0223 Boehringer Ingelheim Investigational Site, Conyers, Georgia
  - 502.373.0268 Boehringer Ingelheim Investigational Site, Sandersville, Georgia
  - 502.373.0245 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 502.373.0199 Boehringer Ingelheim Investigational Site, Tucker, Georgia
  - 502.373.0162 Boehringer Ingelheim Investigational Site, Valdosta, Georgia
  - 502.373.0203 Boehringer Ingelheim Investigational Site, Pocatello, Idaho
  - 502.373.0244 Boehringer Ingelheim Investigational Site, Burbank, Illinois
  - 502.373.0272 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 502.373.0217 Boehringer Ingelheim Investigational Site, Olympia Fields, Illinois
  - 502.373.0270 Boehringer Ingelheim Investigational Site, Des Moines, Iowa
  - 502.373.0167 Boehringer Ingelheim Investigational Site, Monroe, Louisiana
  - 502.373.0158 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 502.373.0247 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 502.373.0284 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 502.373.0229 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 502.373.0237 Boehringer Ingelheim Investigational Site, Wyandotte, Michigan
  - 502.373.0208 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 502.373.0232 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 502.373.0231 Boehringer Ingelheim Investigational Site, Saint Paul, Minnesota
  - 502.373.0181 Boehringer Ingelheim Investigational Site, Biloxi, Mississippi
  - 502.373.0185 Boehringer Ingelheim Investigational Site, Cleveland, Mississippi
  - 502.373.0254 Boehringer Ingelheim Investigational Site, Jackson, Mississippi
  - 502.373.0195 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 502.373.0207 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 502.373.0239 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 502.373.0279 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 502.373.0169 Boehringer Ingelheim Investigational Site, North Las Vegas, Nevada
  - 502.373.0157 Boehringer Ingelheim Investigational Site, Camden, New Jersey
  - 502.373.0202 Boehringer Ingelheim Investigational Site, East Orange, New Jersey
  - 502.373.0191 Boehringer Ingelheim Investigational Site, Newark, New Jersey
  - 502.373.0271 Boehringer Ingelheim Investigational Site, Westwood, New Jersey
  - 502.373.0213 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 502.373.0230 Boehringer Ingelheim Investigational Site, Buffalo, New York
  - 502.373.0288 Boehringer Ingelheim Investigational Site, Kingston, New York
  - 502.373.0238 Boehringer Ingelheim Investigational Site, New York, New York
  - 502.373.0252 Boehringer Ingelheim Investigational Site, New York, New York
  - 502.373.0286 Boehringer Ingelheim Investigational Site, New York, New York
  - 502.373.0166 Boehringer Ingelheim Investigational Site, Northport, New York
  - 502.373.0156 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 502.373.0264 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 502.373.0227 Boehringer Ingelheim Investigational Site, Scarsdale, New York
  - 502.373.0150 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 502.373.0163 Boehringer Ingelheim Investigational Site, Westfield, New York
  - 502.373.0241 Boehringer Ingelheim Investigational Site, Williamsville, New York
  - 502.373.0273 Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - 502.373.0261 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 502.373.0222 Boehringer Ingelheim Investigational Site, Fargo, North Dakota
  - 502.373.0155 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 502.373.0164 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 502.373.0168 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 502.373.0159 Boehringer Ingelheim Investigational Site, Mansfield, Ohio
  - 502.373.0178 Boehringer Ingelheim Investigational Site, Oklahoma City, Ohio
  - 502.373.0259 Boehringer Ingelheim Investigational Site, Guthrie, Oklahoma
  - 502.373.0154 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 502.373.0152 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 502.373.0243 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 502.373.0265 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 502.373.0153 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 502.373.0274 Boehringer Ingelheim Investigational Site, Sellersville, Pennsylvania
  - 502.373.0184 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 502.373.0248 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 502.373.0172 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 502.373.0187 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 502.373.0219 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 502.373.0275 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 502.373.0221 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 502.373.0206 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 502.373.0234 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 502.373.0280 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 502.373.0249 Boehringer Ingelheim Investigational Site, Burke, Virginia
  - 502.373.0281 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 502.373.0212 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Argentina (24):
  - 502.373.350 Boehringer Ingelheim Investigational Site, Capital Federal
  - 502.373.351 Boehringer Ingelheim Investigational Site, Capital Federal
  - 502.373.352 Boehringer Ingelheim Investigational Site, Capital Federal
  - 502.373.353 Boehringer Ingelheim Investigational Site, Capital Federal
  - 502.373.354 Boehringer Ingelheim Investigational Site, Capital Federal
  - 502.373.355 Boehringer Ingelheim Investigational Site, Capital Federal
  - 502.373.356 Boehringer Ingelheim Investigational Site, Capital Federal
  - 502.373.378 Boehringer Ingelheim Investigational Site, Capital Federal
  - 502.373.362 Boehringer Ingelheim Investigational Site, Corones Suárez
  - 502.373.357 Boehringer Ingelheim Investigational Site, Córdoba
  - 502.373.358 Boehringer Ingelheim Investigational Site, Córdoba
  - 502.373.360 Boehringer Ingelheim Investigational Site, Córdoba
  - 502.373.361 Boehringer Ingelheim Investigational Site, Córdoba
  - 502.373.377 Boehringer Ingelheim Investigational Site, Córdoba
  - 502.373.364 Boehringer Ingelheim Investigational Site, La Plata
  - 502.373.365 Boehringer Ingelheim Investigational Site, Mar del Plata
  - 502.373.366 Boehringer Ingelheim Investigational Site, Mendoza
  - 502.373.376 Boehringer Ingelheim Investigational Site, Mendoza
  - 502.373.367 Boehringer Ingelheim Investigational Site, Rosario
  - 502.373.369 Boehringer Ingelheim Investigational Site, Salta
  - 502.373.371 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
  - 502.373.373 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
  - 502.373.375 Boehringer Ingelheim Investigational Site, Santa Fe
  - 502.373.374 Boehringer Ingelheim Investigational Site, Zárate
- Australia (33):
  - 502.373.0534 The Canberra Hospital, Woden, Australian Capital Territory
  - 502.373.0536 Royal Prince Alfred Hospital, Camperdown, New South Wales
  - 502.373.0544 Coffs Harbour Cardiovascular Clinic, Coffs Harbour, New South Wales
  - 502.373.0538 Concord Repatriation General Hospital, Concord, New South Wales
  - 502.373.0539 Central Coast Neuroscience Research, Gosford, New South Wales
  - 502.373.0556 Gosford Hospital, Gosford, New South Wales
  - 502.373.0542 St. George Hospital, Kogarah, New South Wales
  - 502.373.0552 St George Private Hospital, Kogarah, New South Wales
  - 502.373.0559 St George Hospital - Dept of Clinical Pharmacology, Kogarah, New South Wales
  - 502.373.0528 John Hunter Hospital, Newcastle, New South Wales
  - 502.373.0535 The Prince of Wales Hospital, Randwick, New South Wales
  - 502.373.0533 Royal North Shore Hospital, St Leonards, New South Wales
  - 502.373.0549 Illawarra Regional Hospital, Wollongong, New South Wales
  - 502.373.0523 The Prince Charles Hospital, Chermside, Queensland
  - 502.373.0524 Royal Brisbane Hospital, Herston, Queensland
  - 502.373.0526 Peninsula Clinical Research Centre, Kippa-Ring, Queensland
  - 502.373.0540 Gold Coast Hospital, Southport, Queensland
  - 502.373.0521 Princess Alexandra Hospital, Woolloongabba, Queensland
  - 502.373.0546 Flinders Medical Centre, Bedford Park, South Australia
  - 502.373.0550 Repatriation General Hospital, Daw Park, South Australia
  - 502.373.0551 Port Lincoln "The Investigator" Clinic, Port Lincoln, South Australia
  - 502.373.0529 Launceston General Hospital, Launceston, Tasmania
  - 502.373.0531 Box Hill Hospital, Box Hill, Victoria
  - 502.373.0548 The Northern Hospital, Epping, Victoria
  - 502.373.0522 The Geelong Hospital, Geelong, Victoria
  - 502.373.0520 Royal Melbourne Hospital, Parkville, Victoria
  - 502.373.0525 The Alfred Hospital, Prahran, Victoria
  - 502.373.0532 Baker Medical Research Centre, Prahran, Victoria
  - 502.373.0557 Maroondah Hospital, Ringwood East, Victoria
  - 502.373.0537 Austin & Repatriation Medical Centre, West Heidelberg, Victoria
  - 502.373.0547 Fremantle Hospital, Fremantle, Western Australia
  - 502.373.0530 Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - 502.373.0545 Royal Perth Hospital, Perth, Western Australia
- Austria (5):
  - 502.373.1128 Boehringer Ingelheim Investigational Site, Graz
  - 502.373.1126 Boehringer Ingelheim Investigational Site, Vienna
  - 502.373.1127 Boehringer Ingelheim Investigational Site, Vienna
  - 502.373.1129 Boehringer Ingelheim Investigational Site, Vienna
  - 502.373.1125 Boehringer Ingelheim Investigational Site, Wels
- Belgium (20):
  - 502.373.1004 Boehringer Ingelheim Investigational Site, Aalst
  - 502.373.1015 Boehringer Ingelheim Investigational Site, Anderlecht
  - 502.373.1005 Boehringer Ingelheim Investigational Site, Antwerp
  - 502.373.1022 Boehringer Ingelheim Investigational Site, Bornem
  - 502.373.1021 Boehringer Ingelheim Investigational Site, Brasschaat
  - 502.373.1003 Boehringer Ingelheim Investigational Site, Bruges
  - 502.373.1017 Boehringer Ingelheim Investigational Site, Charleroi
  - 502.373.1009 Boehringer Ingelheim Investigational Site, Genk
  - 502.373.1018 Boehringer Ingelheim Investigational Site, Godinne
  - 502.373.1011 Boehringer Ingelheim Investigational Site, Haine-Saint-Paul
  - 502.373.1019 Boehringer Ingelheim Investigational Site, Haine-Saint-Paul
  - 502.373.1007 Boehringer Ingelheim Investigational Site, Hasselt
  - 502.373.1000 Boehringer Ingelheim Investigational Site, Leuven
  - 502.373.1020 Boehringer Ingelheim Investigational Site, Mechelen
  - 502.373.1006 Boehringer Ingelheim Investigational Site, Mol
  - 502.373.1028 Boehringer Ingelheim Investigational Site, Roeselare
  - 502.373.1014 Boehringer Ingelheim Investigational Site, Seraing
  - 502.373.1002 Boehringer Ingelheim Investigational Site, Turnhout
  - 502.373.1010 Boehringer Ingelheim Investigational Site, Turnhout
  - 502.373.1025 Boehringer Ingelheim Investigational Site, Woluwé-Saint-Lambert
- Brazil (26):
  - 502.373.405 Boehringer Ingelheim Investigational Site, Belo Horizonte
  - 502.373.412 Boehringer Ingelheim Investigational Site, Belo Horizonte
  - 502.373.426 Boehringer Ingelheim Investigational Site, Belo Horizonte
  - 502.373.418 Boehringer Ingelheim Investigational Site, Botucatu
  - 502.373.407 Boehringer Ingelheim Investigational Site, Campinas
  - 502.373.419 Boehringer Ingelheim Investigational Site, Campinas
  - 502.373.425 Boehringer Ingelheim Investigational Site, Cerqueira César - São Paulo
  - 502.373.406 Boehringer Ingelheim Investigational Site, Curitiba
  - 502.373.411 Boehringer Ingelheim Investigational Site, Goiânia
  - 502.373.403 Boehringer Ingelheim Investigational Site, Marília
  - 502.373.400 Boehringer Ingelheim Investigational Site, Pelotas
  - 502.373.416 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 502.373.417 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 502.373.415 Boehringer Ingelheim Investigational Site, Porto Alegre - Rs
  - 502.373.420 Boehringer Ingelheim Investigational Site, Ribeirão Preto
  - 502.373.414 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 502.373.413 Boehringer Ingelheim Investigational Site, Rio de Janeiro - Rj
  - 502.373.409 Boehringer Ingelheim Investigational Site, Salvador
  - 502.373.410 Boehringer Ingelheim Investigational Site, Salvador
  - 502.373.404 Boehringer Ingelheim Investigational Site, Santa Catalina
  - 502.373.421 Boehringer Ingelheim Investigational Site, São José do Rio Preto
  - 502.373.402 Boehringer Ingelheim Investigational Site, São Paulo
  - 502.373.408 Boehringer Ingelheim Investigational Site, São Paulo
  - 502.373.422 Boehringer Ingelheim Investigational Site, São Paulo
  - 502.373.424 Boehringer Ingelheim Investigational Site, São Paulo
  - 502.373.423 Boehringer Ingelheim Investigational Site, Vila Clementino, São Paulo
- Canada (74):
  - 502.373.0001 C849 Division of Cardiology, Foothills Medical Centre, Calgary, Alberta
  - 502.373.0071 Peter Lougheed Centre, Calgary, Alberta
  - 502.373.0020 CHA/University Hospital, Edmonton, Alberta
  - 502.373.0073 Alder Medical Centre, Campbell River, British Columbia
  - 502.373.0062 Gain Medical Centre, Coquitlam, British Columbia
  - 502.373.0046 Interior Clinical Research Consultants Ltd, Kelowna, British Columbia
  - 502.373.0038 New West Cardiac Research, New Westminster, British Columbia
  - 502.373.0048 Suite 100, North Vancouver, British Columbia
  - 502.373.0002 Penticton Regional Hospital, Penticton, British Columbia
  - 502.373.0009 Vancouver Hospital, Vancouver, British Columbia
  - 502.373.0003 Discovery Clinical Services Ltd, Victoria, British Columbia
  - 502.373.0030 Portage Clinical Studies, Manitoba, Manitoba
  - 502.373.0050 St. Pierre Medical Clinic, Saint Pierre, Manitoba
  - 502.373.0077 Health Science Centre Diabetes Research Group, Winnipeg, Manitoba
  - 502.373.0005 Dr. Jeffrey Hiscock, St. John's, Newfoundland and Labrador
  - 502.373.0006 The General Hospital, St. John's, Newfoundland and Labrador
  - 502.373.0056 Antigonish Clinical Trials, Antigonish, Nova Scotia
  - 502.373.0045 Queen Elizabeth II HSC, Halifax, Nova Scotia
  - 502.373.0031 Brampton Research Associates, Brampton, Ontario
  - 502.373.0007 Sudbury Cardiac Research, Greater Sudbury, Ontario
  - 502.373.0011 St. Joseph's Hospital Cardiac Research, Hamilton, Ontario
  - 502.373.0034 HGH McMaster Clinic, Hamilton, Ontario
  - 502.373.0035 Hamilton Medical Research, Hamilton, Ontario
  - 502.373.0064 Chedoke Hospital, Hamilton, Ontario
  - 502.373.0082 3U4, McMaster University Medical Centre, Hamilton, Ontario
  - 502.373.0085 HGH McMaster Clinic, Hamilton, Ontario
  - 502.373.0024 London HSC - University Hospital, London, Ontario
  - 502.373.0044 Mississauga Clinical Research Centre, Mississauga, Ontario
  - 502.373.0043 Fraser Clinical Trial Inc, New Westminster, Ontario
  - 502.373.0032 New Market Cardiology Research Grp, Newmarket, Ontario
  - 502.373.0037 Niagara Falls Medical Centre, Niagara Falls, Ontario
  - 502.373.0054 Orleans Medical-Dental Centre, Orléans, Ontario
  - 502.373.0058 Medical Sciences Building, Oshawa, Ontario
  - 502.373.0063 Paradigm Clinical Trials, Oshawa, Ontario
  - 502.373.0029 Riverside Professional Building, Ottawa, Ontario
  - 502.373.0051 Merivale Cardiovascular Consultants, Ottawa, Ontario
  - 502.373.0040 Etobicok Cardiology, Rexdale, Ontario
  - 502.373.0023 Group Health Centre - Clinical Trials, Sault Ste. Marie, Ontario
  - 502.373.0039 Scarborough Cardiology Research, Scarborough Village, Ontario
  - 502.373.0061 CLIKS Medical Research Corp, Thunder Bay, Ontario
  - 502.373.0042 Sunnybrook & Woman's College Health Science Centre, Toronto, Ontario
  - 502.373.0083 St. Michael's Hospital, Toronto, Ontario
  - 502.373.0052 Dr. Bruce Lubelsky, Willowdale, Ontario
  - 502.373.0008 Windsor Health Clinic, Windsor, Ontario
  - 502.373.0081 Centre de recherche clinique, CUSE 3001, Fleurimont, Quebec
  - 502.373.0076 Centre Hospitalier de Vallees de l'Outaouais Gatineau, Gatineau, Quebec
  - 502.373.0057 Centre De Recherche Clinique, Laval, Quebec
  - 502.373.0033 Clinique de Cardiologie de Levis, Lévis, Quebec
  - 502.373.0010 Recherche Invascor, Longueuil, Quebec
  - 502.373.0013 Suite 170, Longueuil, Quebec
  - 502.373.0014 Via Car Recherche Clinique Inc, Longueuil, Quebec
  - 502.373.0015 C/O Peter Carmichael, Longueuil, Quebec
  - 502.373.0016 Suite 170, Longueuil, Quebec
  - 502.373.0017 Suite 170, Longueuil, Quebec
  - 502.373.0086 Via Car Recherche Clinique Inc, Longueuil, Quebec
  - 502.373.0018 Montreal Heart Institute, Montreal, Quebec
  - 502.373.0021 Medi - recherche Inc., Montreal, Quebec
  - 502.373.0022 CHUM - Hotel Dieu, Montreal, Quebec
  - 502.373.0025 Hopital Maisonneuve Rosemont, Montreal, Quebec
  - 502.373.0079 Jewish General Hospital, Montreal, Quebec
  - 502.373.0028 Hop. Du St. Sacrement, Québec, Quebec
  - 502.373.0041 Recherches Clinicar Inc., Québec, Quebec
  - 502.373.0080 Polyclinique vasculaire Centre hospitalier universitaire de, Québec, Quebec
  - 502.373.0084 CHA-Hopital de l'Efant-Jesus, Québec, Quebec
  - 502.373.0027 Ctr Hospitalier Beauce Etchemin, Saint George de Beauce, Quebec
  - 502.373.0012 Hopital Laval - Institute Cardiologie de Quebec, Ste-Foy, Quebec
  - 502.373.0026 Centre hospitalier Pierre-Le Gardeur, Terrebonne, Quebec
  - 502.373.0072 Chra, Thetford-Mines, Quebec
  - 502.373.0053 Mount Royal Clinic, Saskatoon, Saskatchewan
  - 502.373.0055 Specialists - Internal Medicine, Saskatoon, Saskatchewan
  - 502.373.0066 SDRI - University of Saskatchewan, Saskatoon, Saskatchewan
  - 502.373.0067 SDRI - University of Saskatchewan, Saskatoon, Saskatchewan
  - 502.373.0068 SDRI - University of Saskatchewan, Saskatoon, Saskatchewan
  - 502.373.0070 SDRI - University of Saskatchewan, Saskatoon, Saskatchewan
- China (33):
  - 502.373.0601 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0602 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0603 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0604 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0605 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0606 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0607 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0621 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0622 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0623 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0626 Boehringer Ingelheim Investigational Site, Beijing
  - 502.373.0616 Boehringer Ingelheim Investigational Site, Changsha
  - 502.373.0613 Boehringer Ingelheim Investigational Site, Chengdu
  - 502.373.0625 Boehringer Ingelheim Investigational Site, Chengdu
  - 502.373.0620 Boehringer Ingelheim Investigational Site, Guangzhou
  - 502.373.0612 Boehringer Ingelheim Investigational Site, Harbin
  - 502.373.0634 Boehringer Ingelheim Investigational Site, HeBei Province
  - 502.373.0624 Boehringer Ingelheim Investigational Site, Henan Province
  - 502.373.0627 Boehringer Ingelheim Investigational Site, Hubei Province
  - 502.373.0614 Boehringer Ingelheim Investigational Site, Nanjing
  - 502.373.0629 Boehringer Ingelheim Investigational Site, Qingdao
  - 502.373.0632 Boehringer Ingelheim Investigational Site, ShanDong Province
  - 502.373.0633 Boehringer Ingelheim Investigational Site, ShanDong Province
  - 502.373.0617 Boehringer Ingelheim Investigational Site, Shanghai
  - 502.373.0618 Boehringer Ingelheim Investigational Site, Shanghai
  - 502.373.0619 Boehringer Ingelheim Investigational Site, Shanghai
  - 502.373.0628 Boehringer Ingelheim Investigational Site, Shenyang
  - 502.373.0611 Boehringer Ingelheim Investigational Site, Shijiazhuang
  - 502.373.0615 Boehringer Ingelheim Investigational Site, Tianjin
  - 502.373.0631 Boehringer Ingelheim Investigational Site, Tianjin
  - 502.373.0630 Boehringer Ingelheim Investigational Site, Weizikeng
  - 502.373.0608 Boehringer Ingelheim Investigational Site, Wuhan
  - 502.373.0610 Boehringer Ingelheim Investigational Site, Zhenzhou
- Czechia (10):
  - 502.373.1053 Boehringer Ingelheim Investigational Site, Brno
  - 502.373.1060 Boehringer Ingelheim Investigational Site, Havířov
  - 502.373.1055 Boehringer Ingelheim Investigational Site, Kladno
  - 502.373.1059 Boehringer Ingelheim Investigational Site, Mladá Boleslav
  - 502.373.1061 Boehringer Ingelheim Investigational Site, Pilsen
  - 502.373.1051 Boehringer Ingelheim Investigational Site, Prague
  - 502.373.1057 Boehringer Ingelheim Investigational Site, Prague
  - 502.373.1062 Boehringer Ingelheim Investigational Site, Prague
  - 502.373.1056 Boehringer Ingelheim Investigational Site, Příbram
  - 502.373.1058 Boehringer Ingelheim Investigational Site, Ústí nad Orlicí
- Denmark (12):
  - 502.373.1450 Boehringer Ingelheim Investigational Site, Aalborg
  - 502.373.1453 Boehringer Ingelheim Investigational Site, Aarhus C
  - 502.373.1460 Boehringer Ingelheim Investigational Site, Elsinore
  - 502.373.1455 Boehringer Ingelheim Investigational Site, Frederiksberg
  - 502.373.1459 Boehringer Ingelheim Investigational Site, Frederiksberg C
  - 502.373.1458 Boehringer Ingelheim Investigational Site, Hilleroed
  - 502.373.1451 Boehringer Ingelheim Investigational Site, Holbæk
  - 502.373.1452 Boehringer Ingelheim Investigational Site, Hvidovre
  - 502.373.1461 Boehringer Ingelheim Investigational Site, Kjellerup
  - 502.373.1456 Boehringer Ingelheim Investigational Site, Randers
  - 502.373.1457 Boehringer Ingelheim Investigational Site, Slagelse
  - 502.373.1454 Boehringer Ingelheim Investigational Site, Svendborg
- Finland (10):
  - 502.373.1486 Boehringer Ingelheim Investigational Site, Hämeenlinna
  - 502.373.1470 Boehringer Ingelheim Investigational Site, Helsinki
  - 502.373.1473 Boehringer Ingelheim Investigational Site, Helsinki
  - 502.373.1479 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 502.373.1488 Boehringer Ingelheim Investigational Site, Kuopio
  - 502.373.1481 Boehringer Ingelheim Investigational Site, Kuusankoski
  - 502.373.1487 Boehringer Ingelheim Investigational Site, Liperi
  - 502.373.1475 Boehringer Ingelheim Investigational Site, Oulun Kaupunki
  - 502.373.1471 Boehringer Ingelheim Investigational Site, Turku
  - 502.373.1485 Boehringer Ingelheim Investigational Site, Vantaa
- France (25):
  - 502.373.1093 Cabinet Médical, Albens
  - 502.373.1090 Cabinet Médical, Béziers
  - 502.373.1075 Cabinet Médical, Bourges
  - 502.373.1091 Cabinet Médical, Broglie
  - 502.373.1097 Cabinet Médical, Castelnaudary
  - 502.373.1089 Cabinet Médical, Gémenos
  - 502.373.1099 Cabinet Médical, Husseren Wesserlin
  - 502.373.1094 Cabinet Médical, Hyères
  - 502.373.1078 Cabinet Médical des Tanneurs, L'Aigle
  - 502.373.1096 Cabinet Médical, La Rochelle
  - 502.373.1081 Cabinet Médical, Le Pradet
  - 502.373.1083 Cabinet Médical, Mûrs-Erigné
  - 502.373.1084 Cabinet Médical, Nantes
  - 502.373.1086 Cabinet Médical, Nantes
  - 502.373.1080 Cabinet Médical, Niort
  - 502.373.1095 Cabinet Médical, Orthez
  - 502.373.1079 Cabinet Médical, Paris
  - 502.373.1088 Cabinet Médical, Rennes
  - 502.373.1098 Cabinet Médical, Rosiers-d'Égletons
  - 502.373.1076 Cabinet Médical La Grande Ramée, Saint Martin dHyeres
  - 502.373.1085 Cabinet Médical, Saint-Julien-des-Landes
  - 502.373.1092 Cabinet Médical de St Pierre, Saint-Pierre-de-Chandieu
  - 502.373.1077 Cabinet Médical, Saint-Romain-sur-Cher
  - 502.373.1087 Cabinet Médical, Strasbourg
  - 502.373.1082 Cabinet Médical, Tours
- Germany (35):
  - 502.373.1164 Boehringer Ingelheim Investigational Site, Bad Lausick
  - 502.373.1166 Boehringer Ingelheim Investigational Site, Bad Lauterberg im Harz
  - 502.373.1138 Boehringer Ingelheim Investigational Site, Bad Mergentheim
  - 502.373.1156 Boehringer Ingelheim Investigational Site, Berlin
  - 502.373.1160 Boehringer Ingelheim Investigational Site, Berlin
  - 502.373.1161 Boehringer Ingelheim Investigational Site, Berlin
  - 502.373.1144 Boehringer Ingelheim Investigational Site, Bielefeld
  - 502.373.1137 Boehringer Ingelheim Investigational Site, Cologne
  - 502.373.1152 Boehringer Ingelheim Investigational Site, Dessau
  - 502.373.1139 Boehringer Ingelheim Investigational Site, Dortmund
  - 502.373.1159 Boehringer Ingelheim Investigational Site, Dortmund
  - 502.373.1136 Boehringer Ingelheim Investigational Site, Dresden
  - 502.373.1145 Boehringer Ingelheim Investigational Site, Eberswalde
  - 502.373.1155 Boehringer Ingelheim Investigational Site, Erlangen
  - 502.373.1157 Boehringer Ingelheim Investigational Site, Essen
  - 502.373.1153 Boehringer Ingelheim Investigational Site, Haag
  - 502.373.1148 Boehringer Ingelheim Investigational Site, Hamburg
  - 502.373.1132 Boehringer Ingelheim Investigational Site, Heidelberg
  - 502.373.1131 Boehringer Ingelheim Investigational Site, Homburg/Saar
  - 502.373.1147 Boehringer Ingelheim Investigational Site, Karlsburg
  - 502.373.1154 Boehringer Ingelheim Investigational Site, Kelkheim
  - 502.373.1142 Boehringer Ingelheim Investigational Site, Künzing
  - 502.373.1165 Boehringer Ingelheim Investigational Site, Lübeck
  - 502.373.1134 Boehringer Ingelheim Investigational Site, Mainz
  - 502.373.1133 Boehringer Ingelheim Investigational Site, Melsungen
  - 502.373.1146 Boehringer Ingelheim Investigational Site, München
  - 502.373.1149 Boehringer Ingelheim Investigational Site, Offenbach
  - 502.373.1162 Boehringer Ingelheim Investigational Site, Riesa
  - 502.373.1140 Boehringer Ingelheim Investigational Site, Rostock
  - 502.373.1150 Boehringer Ingelheim Investigational Site, Sindelfingen
  - 502.373.1163 Boehringer Ingelheim Investigational Site, Starnberg
  - 502.373.1158 Boehringer Ingelheim Investigational Site, Stuttgart
  - 502.373.1167 Boehringer Ingelheim Investigational Site, Timmendorfer Strand
  - 502.373.1135 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 502.373.1141 Boehringer Ingelheim Investigational Site, Witten
- Greece (15):
  - 502.373.1200 Boehringer Ingelheim Investigational Site, Athens
  - 502.373.1203 Boehringer Ingelheim Investigational Site, Athens
  - 502.373.1206 Boehringer Ingelheim Investigational Site, Athens
  - 502.373.1207 Boehringer Ingelheim Investigational Site, Athens
  - 502.373.1208 Boehringer Ingelheim Investigational Site, Athens
  - 502.373.1214 Boehringer Ingelheim Investigational Site, Athens
  - 502.373.1224 Boehringer Ingelheim Investigational Site, Corinth
  - 502.373.1209 Boehringer Ingelheim Investigational Site, Elefsina
  - 502.373.1211 Boehringer Ingelheim Investigational Site, Goudi/ Athens
  - 502.373.1201 Boehringer Ingelheim Investigational Site, Ioannina
  - 502.373.1210 Boehringer Ingelheim Investigational Site, Kavala,greece
  - 502.373.1202 Boehringer Ingelheim Investigational Site, Melissia, Athens
  - 502.373.1205 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 502.373.1213 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 502.373.1204 Boehringer Ingelheim Investigational Site, Véria
- Hong Kong (5):
  - 502.373.0676 Boehringer Ingelheim Investigational Site, Hong Kong
  - 502.373.0677 Boehringer Ingelheim Investigational Site, Hong Kong
  - 502.373.0680 Boehringer Ingelheim Investigational Site, Hong Kong
  - 502.373.0681 Boehringer Ingelheim Investigational Site, Hong Kong
  - 502.373.0685 Boehringer Ingelheim Investigational Site, Hong Kong
- Hungary (20):
  - 502.373.1227 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1230 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1231 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1232 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1233 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1235 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1237 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1239 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1242 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1244 Boehringer Ingelheim Investigational Site, Budapest
  - 502.373.1236 Boehringer Ingelheim Investigational Site, Debrecen
  - 502.373.1240 Boehringer Ingelheim Investigational Site, Debrecen
  - 502.373.1228 Boehringer Ingelheim Investigational Site, Kecskemét
  - 502.373.1241 Boehringer Ingelheim Investigational Site, Nyíregyháza
  - 502.373.1226 Boehringer Ingelheim Investigational Site, Pécs
  - 502.373.1229 Boehringer Ingelheim Investigational Site, Siófok
  - 502.373.1238 Boehringer Ingelheim Investigational Site, Szeged
  - 502.373.1225 Boehringer Ingelheim Investigational Site, Székesfehérvár
  - 502.373.1234 Boehringer Ingelheim Investigational Site, Tatabánya
  - 502.373.1243 Boehringer Ingelheim Investigational Site, Veszprém
- Ireland (4):
  - 502.373.1714 Dept. of Clinical Pharmacology, Dublin
  - 502.373.1717 Adelaide & Meath Hospitals, Dublin
  - 502.373.1719 Pulmonary Function Laboratory, Dublin
  - 502.373.1720 Mallow General Hospital, Mallow
- Italy (30):
  - 502.373.1257 Ospedale "Mazzoni", Ascoli Piceno
  - 502.373.1259 Ospedale di Bentivoglio, Bentivoglio (BO)
  - 502.373.1255 Ospedale "S. Orsola Malpighi", Bologna
  - 502.373.1278 Ospedale Bellaria, Bologna
  - 502.373.1275 A.O. Spedali Civili di Brescia -Univ. degli studi di Brescia, Brescia
  - 502.373.1261 Ospedale Civile di Casarano, Casarano (LE)
  - 502.373.1252 Azienda Ospedaliera di Caserta, Caserta
  - 502.373.1254 Ospedale di Città della Pieve, Città Della Pieve (PG)
  - 502.373.1262 Arcispedale "S. Anna", Ferrara
  - 502.373.1250 Ospedale Civile "S. Polo", Monfalcone (go)
  - 502.373.1266 Azienda Universitaria Policlinico "Federico II", Napoli
  - 502.373.1267 Azienda Universitaria Policlinico II, Napoli
  - 502.373.1269 Università Federico II, Napoli
  - 502.373.1279 Asl Na 1, Napoli
  - 502.373.1264 Presidio Ospedaliero "Villa Sofia", Palermo
  - 502.373.1265 IRCCS - Policlinico S. Matteo, Pavia
  - 502.373.1251 Policlinico Monteluce, Perugia
  - 502.373.1258 Ospedale "R. Silvestrini", Perugia
  - 502.373.1274 Ospedale "R. Silvestrini", Perugia
  - 502.373.1253 Istituto di Ricovero a Carattere Scientifico Neuromed- IRCCS, Pozzilli (IS)
  - 502.373.1263 Policlinico Umberto I, Roma
  - 502.373.1268 Ospedale "S. Spirito", Roma
  - 502.373.1270 Policlinico di Tor Vergata, Roma
  - 502.373.1273 A.O. "S. Camillo de Lellis", Roma
  - 502.373.1260 Ospedale "N. Melli", S. Pietro Vernotico (BR)
  - 502.373.1256 Ospedale Civile SS. Annunziata - USL 1, Sassari
  - 502.373.1277 A.S.O. "S. Giovanni Battista", Torino
  - 502.373.1272 Ospedale di Circolo di Varese, Varese
  - 502.373.1271 Ospedale Civile, Venezia
  - 502.373.1276 Ospedale Belcolle, Viterbo
- Malaysia (8):
  - 502.373.0733 Boehringer Ingelheim Investigational Site, George Town
  - 502.373.0736 Boehringer Ingelheim Investigational Site, Johor Bahru
  - 502.373.2707 Boehringer Ingelheim Investigational Site, Kelantan Darul Naim
  - 502.373.0739 Boehringer Ingelheim Investigational Site, Kelantan
  - 502.373.0732 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 502.373.0734 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 502.373.60001 Boehringer Ingelheim Investigational Site, Kuala Selangor
  - 502.373.0731 Boehringer Ingelheim Investigational Site, Putrajaya
- Mexico (12):
  - 502.373.0450 Boehringer Ingelheim Investigational Site, Guadalajara
  - 502.373.0451 Boehringer Ingelheim Investigational Site, Guadalajara
  - 502.373.0452 Boehringer Ingelheim Investigational Site, Guadalajara
  - 502.373.0459 Boehringer Ingelheim Investigational Site, Guadalajara
  - 502.373.0460 Boehringer Ingelheim Investigational Site, Guadalajara
  - 502.373.0461 Boehringer Ingelheim Investigational Site, Guadalajara
  - 502.373.0470 Boehringer Ingelheim Investigational Site, Guadalajara
  - 502.373.0457 Boehringer Ingelheim Investigational Site, México
  - 502.373.0458 Boehringer Ingelheim Investigational Site, México
  - 502.373.0454 Boehringer Ingelheim Investigational Site, Monterrey
  - 502.373.0453 Boehringer Ingelheim Investigational Site, Zapopan
  - 502.373.0456 Boehringer Ingelheim Investigational Site, Zapopan
- Netherlands (23):
  - 502.373.1313 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 502.373.1309 Boehringer Ingelheim Investigational Site, Amsterdam
  - 502.373.1305 Boehringer Ingelheim Investigational Site, Beverwijk
  - 502.373.1302 Boehringer Ingelheim Investigational Site, Doetinchem
  - 502.373.1304 Boehringer Ingelheim Investigational Site, Drachten
  - 502.373.1301 Boehringer Ingelheim Investigational Site, Eindhoven
  - 502.373.1318 Boehringer Ingelheim Investigational Site, Ermelo
  - 502.373.1320 Boehringer Ingelheim Investigational Site, Ewijk
  - 502.373.1310 Boehringer Ingelheim Investigational Site, Hengelo
  - 502.373.1303 Boehringer Ingelheim Investigational Site, Hoorn
  - 502.373.1322 Boehringer Ingelheim Investigational Site, Huizen
  - 502.373.1300 Boehringer Ingelheim Investigational Site, Lichtenvoorde
  - 502.373.1323 Boehringer Ingelheim Investigational Site, Losser
  - 502.373.1307 Boehringer Ingelheim Investigational Site, Nieuwegein
  - 502.373.1317 Boehringer Ingelheim Investigational Site, Rijswijk
  - 502.373.1319 Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - 502.373.1308 Boehringer Ingelheim Investigational Site, Rotterdam
  - 502.373.1321 Boehringer Ingelheim Investigational Site, Spijkenisse
  - 502.373.1311 Boehringer Ingelheim Investigational Site, Stadskanaal
  - 502.373.1312 Boehringer Ingelheim Investigational Site, The Hague
  - 502.373.1314 Boehringer Ingelheim Investigational Site, Tilburg
  - 502.373.1316 Boehringer Ingelheim Investigational Site, Utrecht
  - 502.373.1315 Boehringer Ingelheim Investigational Site, Velp
- New Zealand (8):
  - 502.373.0500 Boehringer Ingelheim Investigational Site, Auckland
  - 502.373.0502 Boehringer Ingelheim Investigational Site, Auckland
  - 502.373.0507 Boehringer Ingelheim Investigational Site, Christchurch
  - 502.373.0504 Boehringer Ingelheim Investigational Site, Hamiton
  - 502.373.0506 Boehringer Ingelheim Investigational Site, Hasting
  - 502.373.0501 Middlemore Hospital, Otahuhu Auckland
  - 502.373.0503 Boehringer Ingelheim Investigational Site, Takapuna Auckland
  - 502.373.0505 Tauranga Study Centre, Tauranga
- Norway (5):
  - 502.373.20003 Boehringer Ingelheim Investigational Site, Fevik
  - 502.373.20004 Fana Hjertesenter, Nesttun
  - 502.373.20001 Stavanger Universitetssykehus, Stavanger
  - 502.373.20002 Tvedestrand Legesenter, Tvedestrand
  - 502.373.20005 Sykehuset i Vestfold, Avd. Tønsberg, Tønsberg
- Philippines (6):
  - 502.373.0702 De La Salle University Medical Center, Cavite
  - 502.373.0700 Philippine General Hospital, Manila
  - 502.373.0701 Manila Doctors Hospital, Room 3 Annex, Manila
  - 502.373.0705 The Medical City, Pasig
  - 502.373.0703 Philippine Heart Center, Quezon City
  - 502.373.0704 National Kidney & Transplant Institute, Room 821, Quezon City
- Poland (25):
  - 502.373.1354 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 502.373.1366 Boehringer Ingelheim Investigational Site, Częstochowa
  - 502.373.1368 Boehringer Ingelheim Investigational Site, Gdynia
  - 502.373.1365 Boehringer Ingelheim Investigational Site, Gdynia Redlowo
  - 502.373.1359 Boehringer Ingelheim Investigational Site, Grójec
  - 502.373.1369 Boehringer Ingelheim Investigational Site, Grudziądz
  - 502.373.1375 Boehringer Ingelheim Investigational Site, Inowrocław
  - 502.373.1360 Boehringer Ingelheim Investigational Site, Jarosławiec
  - 502.373.1372 Boehringer Ingelheim Investigational Site, Katowice
  - 502.373.1376 Boehringer Ingelheim Investigational Site, Katowice
  - 502.373.1361 Boehringer Ingelheim Investigational Site, Kielce
  - 502.373.1358 Boehringer Ingelheim Investigational Site, Lodz
  - 502.373.1364 Boehringer Ingelheim Investigational Site, Lubartów
  - 502.373.1374 Boehringer Ingelheim Investigational Site, Lubin
  - 502.373.1367 Boehringer Ingelheim Investigational Site, Nowy Sącz
  - 502.373.1356 Boehringer Ingelheim Investigational Site, Piotrkow Trybunalski
  - 502.373.1370 Boehringer Ingelheim Investigational Site, Poznan
  - 502.373.1357 Boehringer Ingelheim Investigational Site, Ruda Śląska
  - 502.373.1352 Boehringer Ingelheim Investigational Site, Skierniewice
  - 502.373.1362 Boehringer Ingelheim Investigational Site, Tarnów
  - 502.373.1355 Boehringer Ingelheim Investigational Site, Tomaszów Mazowiecki
  - 502.373.1353 Boehringer Ingelheim Investigational Site, Torun
  - 502.373.1351 Boehringer Ingelheim Investigational Site, Warsaw
  - 502.373.1363 Boehringer Ingelheim Investigational Site, Warsaw
  - 502.373.1373 Boehringer Ingelheim Investigational Site, Węgrów
- Portugal (10):
  - 502.373.1402 Hospital Garcia de Orta, Almada
  - 502.373.1400 Hospital Fernando Fonseca, Amadora
  - 502.373.1411 Hospital de Santa Cruz, Carnaxide
  - 502.373.1408 Hospitais da Universidade de Coimbra, Coimbra
  - 502.373.1406 Hospital Distrital de Faro Geral, Faro
  - 502.373.1403 Hospital de Santa Marta, Lisbon
  - 502.373.1409 Hospital de Santa Maria, Lisbon
  - 502.373.1401 Unidade Local de Saúde de Matosinhos, Matosinhos Municipality
  - 502.373.1410 Hospital de Santo António, Porto
  - 502.373.1407 Centro Hospitalar vila Nova de Gaia, Vila Nova de Gaia
- Puerto Rico (5):
  - 502.373.0215 Boehringer Ingelheim Investigational Site, Caguas
  - 502.373.0267 Boehringer Ingelheim Investigational Site, Las Lomas
  - 502.373.0190 Boehringer Ingelheim Investigational Site, Manatí
  - 502.373.0198 Boehringer Ingelheim Investigational Site, Orocovis
  - 502.373.0262 Boehringer Ingelheim Investigational Site, Rio Piedras
- Russia (9):
  - 502.373.1425 Boehringer Ingelheim Investigational Site, Moscow
  - 502.373.1426 Boehringer Ingelheim Investigational Site, Moscow
  - 502.373.1427 Boehringer Ingelheim Investigational Site, Moscow
  - 502.373.1428 Boehringer Ingelheim Investigational Site, Moscow
  - 502.373.1429 Boehringer Ingelheim Investigational Site, Moscow
  - 502.373.1430 Boehringer Ingelheim Investigational Site, Moscow
  - 502.373.1433 Boehringer Ingelheim Investigational Site, Moscow
  - 502.373.1431 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 502.373.1432 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Singapore (3):
  - 502.373.2706 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 502.373.0725 Boehringer Ingelheim Investigational Site, Singapore
  - 502.373.0726 Boehringer Ingelheim Investigational Site, Singapore
- Slovakia (5):
  - 502.373.1535 Boehringer Ingelheim Investigational Site, Bratislava
  - 502.373.1529 Boehringer Ingelheim Investigational Site, Košice
  - 502.373.1540 Boehringer Ingelheim Investigational Site, Košice
  - 502.373.1538 Boehringer Ingelheim Investigational Site, Nitra
  - 502.373.1545 Boehringer Ingelheim Investigational Site, Rimavská Sobota
- South Africa (15):
  - 502.373.1553 Boehringer Ingelheim Investigational Site, Bellville
  - 502.373.1552 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 502.373.1550 Boehringer Ingelheim Investigational Site, Cape Town
  - 502.373.1561 Boehringer Ingelheim Investigational Site, Cape Town
  - 502.373.1551 Boehringer Ingelheim Investigational Site, Durban
  - 502.373.1560 Boehringer Ingelheim Investigational Site, Fiachrdtpark, Bloemfontein
  - 502.373.1563 Boehringer Ingelheim Investigational Site, George East
  - 502.373.1554 Boehringer Ingelheim Investigational Site, KwaKhangela
  - 502.373.1555 Boehringer Ingelheim Investigational Site, Park Town West
  - 502.373.1559 Boehringer Ingelheim Investigational Site, Port Elizabeth
  - 502.373.1562 Boehringer Ingelheim Investigational Site, Port Elizabeth
  - 502.373.1558 Boehringer Ingelheim Investigational Site, Soweto
  - 502.373.1557 Boehringer Ingelheim Investigational Site, Sunninghill
  - 502.373.1564 Boehringer Ingelheim Investigational Site, Sunninghill
  - 502.373.1556 Boehringer Ingelheim Investigational Site, Vanderbijlpark
- South Korea (10):
  - 502.373.0763 Boehringer Ingelheim Investigational Site, Incheon
  - 502.373.0764 Boehringer Ingelheim Investigational Site, Kwangju
  - 502.373.0755 Boehringer Ingelheim Investigational Site, Pusan
  - 502.373.0750 Boehringer Ingelheim Investigational Site, Seoul
  - 502.373.0753 Boehringer Ingelheim Investigational Site, Seoul
  - 502.373.0756 Boehringer Ingelheim Investigational Site, Seoul
  - 502.373.0757 Boehringer Ingelheim Investigational Site, Seoul
  - 502.373.0760 Boehringer Ingelheim Investigational Site, Seoul
  - 502.373.0761 Boehringer Ingelheim Investigational Site, Seoul
  - 502.373.0754 Boehringer Ingelheim Investigational Site, Taegu
- Spain (23):
  - 502.373.1582 Boehringer Ingelheim Investigational Site, Alcorcón (Madrid)
  - 502.373.1601 Boehringer Ingelheim Investigational Site, Alicante
  - 502.373.1586 Boehringer Ingelheim Investigational Site, Barcelona
  - 502.373.1590 Boehringer Ingelheim Investigational Site, Barcelona
  - 502.373.1597 Boehringer Ingelheim Investigational Site, Barcelona
  - 502.373.1599 Boehringer Ingelheim Investigational Site, Barcelona
  - 502.373.1595 Boehringer Ingelheim Investigational Site, Burjasot (Valencia)
  - 502.373.1584 Boehringer Ingelheim Investigational Site, Granada
  - 502.373.1585 Boehringer Ingelheim Investigational Site, Granada
  - 502.373.1576 Boehringer Ingelheim Investigational Site, Madrid
  - 502.373.1578 Boehringer Ingelheim Investigational Site, Madrid
  - 502.373.1580 Boehringer Ingelheim Investigational Site, Madrid
  - 502.373.1589 Boehringer Ingelheim Investigational Site, Madrid
  - 502.373.1592 Boehringer Ingelheim Investigational Site, Madrid
  - 502.373.1577 Boehringer Ingelheim Investigational Site, Málaga
  - 502.373.1596 Boehringer Ingelheim Investigational Site, Málaga
  - 502.373.1594 Boehringer Ingelheim Investigational Site, Murcia
  - 502.373.1579 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 502.373.1593 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 502.373.1598 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 502.373.1583 Boehringer Ingelheim Investigational Site, Seville
  - 502.373.1575 Boehringer Ingelheim Investigational Site, Valencia
  - 502.373.1591 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (12):
  - 502.373.1504 Capio Lundby sjukhus, Gothenburg
  - 502.373.1509 Hjärtsektionen / Med.kliniken, Gothenburg
  - 502.373.1514 Hjärt/Kärlforskn.enheten, Gothenburg
  - 502.373.1501 Hjaertmottagningen, Helsingborg
  - 502.373.1505 Jakobsbergs sjukhus, Järfälla
  - 502.373.1502 Borgmästargaardens Läkarmottagning, Malmo
  - 502.373.1506 Hjärtmottagningen, Malmo
  - 502.373.1507 Kardiologiska kliniken, Malmo
  - 502.373.1508 Kolgahuset Läkargrupp, Malmo
  - 502.373.1511 Sjuntorps Vaardcentral, Sjuntorp
  - 502.373.1503 Källtorps Vaardcentral, Trollhättan
  - 502.373.1512 Vännäs Vaardcentral, Vännäs
- Switzerland (10):
  - 502.373.1625 Boehringer Ingelheim Investigational Site, Basel
  - 502.373.1632 Boehringer Ingelheim Investigational Site, Bellinzona
  - 502.373.1634 Boehringer Ingelheim Investigational Site, Bern
  - 502.373.1627 Boehringer Ingelheim Investigational Site, Biel/Bienne
  - 502.373.1631 Boehringer Ingelheim Investigational Site, Chur
  - 502.373.1633 Boehringer Ingelheim Investigational Site, Kreuzlingen
  - 502.373.1639 Boehringer Ingelheim Investigational Site, Lausanne
  - 502.373.1629 Boehringer Ingelheim Investigational Site, Lugano
  - 502.373.1628 Boehringer Ingelheim Investigational Site, Sankt Gallen
  - 502.373.1637 Boehringer Ingelheim Investigational Site, Zurich
- Taiwan (9):
  - 502.373.0780 Boehringer Ingelheim Investigational Site, Changhua
  - 502.373.0779 Boehringer Ingelheim Investigational Site, Chiayi City
  - 502.373.0783 Boehringer Ingelheim Investigational Site, Hualien City
  - 502.373.0776 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 502.373.0778 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 502.373.0775 Boehringer Ingelheim Investigational Site, Tainan
  - 502.373.0777 Boehringer Ingelheim Investigational Site, Tainan
  - 502.373.0781 Boehringer Ingelheim Investigational Site, Taipei
  - 502.373.0782 Boehringer Ingelheim Investigational Site, Taipei
- Thailand (8):
  - 502.373.0801 Boehringer Ingelheim Investigational Site, Bangkok
  - 502.373.0802 Boehringer Ingelheim Investigational Site, Bangkok
  - 502.373.0804 Boehringer Ingelheim Investigational Site, Bangkok
  - 502.373.0805 Boehringer Ingelheim Investigational Site, Bangkok
  - 502.373.0806 Boehringer Ingelheim Investigational Site, Bangkok
  - 502.373.0808 Boehringer Ingelheim Investigational Site, Bangkok
  - 502.373.0803 Boehringer Ingelheim Investigational Site, Khon Kaen
  - 502.373.0807 Boehringer Ingelheim Investigational Site, Nonthaburi
- Turkey (Türkiye) (10):
  - 502.373.1651 Cukurova Universitesi Tip Fakultesi, Adana
  - 502.373.1652 Cukurova Universitesi Tip Fakultesi, Adana
  - 502.373.1653 Ankara Hastanesi Endokrinoloji Bölümü, Ankara
  - 502.373.1656 Baskent Universitesi Tip Fakultesi, Ankara
  - 502.373.1659 Ankara Universitesi Tip Fakultesi, Ankara
  - 502.373.1654 Göztepe SSK Egitim ve Arastirma Hastanesi, Istanbul
  - 502.373.1655 Cerrahpasa Universitesi Tip Fakultesi, Istanbul
  - 502.373.1657 Haseki Hastanesi, Istanbul
  - 502.373.1658 Ege Universitesi Tip Fakultesi, Izmir
  - 502.373.1650 Erciyes Universitesi Tip Fakultesi Kardiyoloji Anabilim Dali, Kayseri
- Ukraine (10):
  - 502.373.1730 Boehringer Ingelheim Investigational Site, Dnyepropetrovsk
  - 502.373.1731 Boehringer Ingelheim Investigational Site, Dnyepropetrovsk
  - 502.373.1728 Boehringer Ingelheim Investigational Site, Kharkiv
  - 502.373.1732 Boehringer Ingelheim Investigational Site, Kharkiv
  - 502.373.1733 Boehringer Ingelheim Investigational Site, Kharkiv
  - 502.373.1725 Boehringer Ingelheim Investigational Site, Kiev
  - 502.373.1726 Boehringer Ingelheim Investigational Site, Kiev
  - 502.373.1727 Boehringer Ingelheim Investigational Site, Kiev
  - 502.373.1729 Boehringer Ingelheim Investigational Site, Kiev
  - 502.373.1734 Boehringer Ingelheim Investigational Site, Kiev
- United Arab Emirates (4):
  - 502.373.1680 Boehringer Ingelheim Investigational Site, Abu Dhabi
  - 502.373.1675 Boehringer Ingelheim Investigational Site, Dubai
  - 502.373.1679 Boehringer Ingelheim Investigational Site, Dubai
  - 502.373.1677 Boehringer Ingelheim Investigational Site, Sharjah city
- United Kingdom (21):
  - 502.373.1698 Boehringer Ingelheim Investigational Site, Aberdeen
  - 502.373.1706 Boehringer Ingelheim Investigational Site, Bathampton
  - 502.373.1690 Boehringer Ingelheim Investigational Site, Belfast
  - 502.373.1694 Boehringer Ingelheim Investigational Site, Birmingham
  - 502.373.1707 Boehringer Ingelheim Investigational Site, Brighton
  - 502.373.1703 Boehringer Ingelheim Investigational Site, Cardiff
  - 502.373.1709 Boehringer Ingelheim Investigational Site, Chichester
  - 502.373.1701 Boehringer Ingelheim Investigational Site, Derby
  - 502.373.1705 Boehringer Ingelheim Investigational Site, Gateshead
  - 502.373.1710 Boehringer Ingelheim Investigational Site, Glasgow
  - 502.373.1700 Boehringer Ingelheim Investigational Site, Kirkcaldy, Fife
  - 502.373.1691 Boehringer Ingelheim Investigational Site, Leeds
  - 502.373.1699 Boehringer Ingelheim Investigational Site, Leicester
  - 502.373.1702 Boehringer Ingelheim Investigational Site, Lincoln
  - 502.373.1697 Boehringer Ingelheim Investigational Site, Liverpool
  - 502.373.1695 Boehringer Ingelheim Investigational Site, London
  - 502.373.1693 Boehringer Ingelheim Investigational Site, Manchester
  - 502.373.1708 Boehringer Ingelheim Investigational Site, Portadown, County Atrim
  - 502.373.1692 Boehringer Ingelheim Investigational Site, Rugby
  - 502.373.1696 Boehringer Ingelheim Investigational Site, Sheffield
  - 502.373.1704 Boehringer Ingelheim Investigational Site, Stirling

REFERENCES:
- [Derived] Lee SF, Ramasundarahettige C, Gerstein HC, McIntyre WF, Eikelboom J, O'Donnell MJ, Zhou Y, Bangdiwala SI, Thabane L. Comparison of total event analysis and first event analysis in relation to heterogeneity in cardiovascular trials. BMC Med Res Methodol. 2025 Jun 9;25(1):159. doi: 10.1186/s12874-025-02593-3. PMID 40490702
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Haring B, Schumacher H, Mancia G, Teo KK, Lonn EM, Mahfoud F, Schmieder R, Mann JFE, Sliwa K, Yusuf S, Bohm M. Triglyceride-glucose index, low-density lipoprotein levels, and cardiovascular outcomes in chronic stable cardiovascular disease: results from the ONTARGET and TRANSCEND trials. Eur J Prev Cardiol. 2024 Feb 15;31(3):311-319. doi: 10.1093/eurjpc/zwad340. PMID 37890035
- [Derived] Cooper TE, Teng C, Tunnicliffe DJ, Cashmore BA, Strippoli GF. Angiotensin-converting enzyme inhibitors and angiotensin receptor blockers for adults with early (stage 1 to 3) non-diabetic chronic kidney disease. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD007751. doi: 10.1002/14651858.CD007751.pub3. PMID 37466151
- [Derived] Bohm M, Schumacher H, Werner C, Teo KK, Lonn EM, Mahfoud F, Speer T, Mancia G, Redon J, Schmieder RE, Sliwa K, Marx N, Weber MA, Laufs U, Williams B, Yusuf S, Mann JFE. Association between exercise frequency with renal and cardiovascular outcomes in diabetic and non-diabetic individuals at high cardiovascular risk. Cardiovasc Diabetol. 2022 Jan 20;21(1):12. doi: 10.1186/s12933-021-01429-w. PMID 35057807
- [Derived] Bohm M, Schumacher H, Teo KK, Lonn EM, Lauder L, Mancia G, Redon J, Schmieder RE, Sliwa K, Marx N, Weber MA, Williams B, Yusuf S, Mann JFE, Mahfoud F. Cardiovascular outcomes in patients at high cardiovascular risk with previous myocardial infarction or stroke. J Hypertens. 2021 Aug 1;39(8):1602-1610. doi: 10.1097/HJH.0000000000002822. PMID 34188004
- [Derived] Bohm M, Schumacher H, Teo KK, Lonn EM, Mahfoud F, Emrich I, Mancia G, Redon J, Schmieder RE, Sliwa K, Lehrke M, Marx N, Weber MA, Williams B, Yusuf S, Mann JFE. Renal outcomes and blood pressure patterns in diabetic and nondiabetic individuals at high cardiovascular risk. J Hypertens. 2021 Apr 1;39(4):766-774. doi: 10.1097/HJH.0000000000002697. PMID 33560052
- [Derived] Mancia G, Schumacher H, Bohm M, Mann JFE, Redon J, Facchetti R, Schmieder RE, Lonn EM, Teo KK, Yusuf S. Visit-to-visit blood pressure variability and renal outcomes: results from ONTARGET and TRANSCEND trials. J Hypertens. 2020 Oct;38(10):2050-2058. doi: 10.1097/HJH.0000000000002567. PMID 32890282
- [Derived] Dehghan M, Mente A, Rangarajan S, Mohan V, Lear S, Swaminathan S, Wielgosz A, Seron P, Avezum A, Lopez-Jaramillo P, Turbide G, Chifamba J, AlHabib KF, Mohammadifard N, Szuba A, Khatib R, Altuntas Y, Liu X, Iqbal R, Rosengren A, Yusuf R, Smuts M, Yusufali A, Li N, Diaz R, Yusoff K, Kaur M, Soman B, Ismail N, Gupta R, Dans A, Sheridan P, Teo K, Anand SS, Yusuf S. Association of egg intake with blood lipids, cardiovascular disease, and mortality in 177,000 people in 50 countries. Am J Clin Nutr. 2020 Apr 1;111(4):795-803. doi: 10.1093/ajcn/nqz348. PMID 31965140
- [Derived] Bohm M, Schumacher H, Teo KK, Lonn EM, Mahfoud F, Mann JFE, Mancia G, Redon J, Schmieder RE, Marx N, Sliwa K, Weber MA, Williams B, Yusuf S. Cardiovascular outcomes and achieved blood pressure in patients with and without diabetes at high cardiovascular risk. Eur Heart J. 2019 Jul 1;40(25):2032-2043. doi: 10.1093/eurheartj/ehz149. PMID 30919899
- [Derived] Bohm M, Schumacher H, Teo KK, Lonn EM, Mahfoud F, Ukena C, Mann JFE, Mancia G, Redon J, Schmieder RE, Sliwa K, Marx N, Weber MA, Williams B, Yusuf S. Resting heart rate and cardiovascular outcomes in diabetic and non-diabetic individuals at high cardiovascular risk analysis from the ONTARGET/TRANSCEND trials. Eur Heart J. 2020 Jan 7;41(2):231-238. doi: 10.1093/eurheartj/ehy808. PMID 30590564
- [Derived] Bohm M, Schumacher H, Teo KK, Lonn EM, Mahfoud F, Mann JFE, Mancia G, Redon J, Schmieder RE, Sliwa K, Weber MA, Williams B, Yusuf S. Achieved blood pressure and cardiovascular outcomes in high-risk patients: results from ONTARGET and TRANSCEND trials. Lancet. 2017 Jun 3;389(10085):2226-2237. doi: 10.1016/S0140-6736(17)30754-7. Epub 2017 Apr 5. PMID 28390695
- [Derived] Dunkler D, Kohl M, Teo KK, Heinze G, Dehghan M, Clase CM, Gao P, Yusuf S, Mann JF, Oberbauer R. Dietary risk factors for incidence or progression of chronic kidney disease in individuals with type 2 diabetes in the European Union. Nephrol Dial Transplant. 2015 Aug;30 Suppl 4:iv76-85. doi: 10.1093/ndt/gfv086. PMID 26209742
- [Derived] Bohm M, Schumacher H, Leong D, Mancia G, Unger T, Schmieder R, Custodis F, Diener HC, Laufs U, Lonn E, Sliwa K, Teo K, Fagard R, Redon J, Sleight P, Anderson C, O'Donnell M, Yusuf S. Systolic blood pressure variation and mean heart rate is associated with cognitive dysfunction in patients with high cardiovascular risk. Hypertension. 2015 Mar;65(3):651-61. doi: 10.1161/HYPERTENSIONAHA.114.04568. Epub 2015 Jan 12. PMID 25583157
- [Derived] Verdecchia P, Reboldi G, Angeli F, Trimarco B, Mancia G, Pogue J, Gao P, Sleight P, Teo K, Yusuf S. Systolic and diastolic blood pressure changes in relation with myocardial infarction and stroke in patients with coronary artery disease. Hypertension. 2015 Jan;65(1):108-14. doi: 10.1161/HYPERTENSIONAHA.114.04310. Epub 2014 Oct 20. PMID 25331850
- [Derived] Lonn EM, Rambihar S, Gao P, Custodis FF, Sliwa K, Teo KK, Yusuf S, Bohm M. Heart rate is associated with increased risk of major cardiovascular events, cardiovascular and all-cause death in patients with stable chronic cardiovascular disease: an analysis of ONTARGET/TRANSCEND. Clin Res Cardiol. 2014 Feb;103(2):149-59. doi: 10.1007/s00392-013-0644-4. Epub 2013 Dec 20. PMID 24356937
- [Derived] Heerspink HJ, Gao P, de Zeeuw D, Clase C, Dagenais GR, Sleight P, Lonn E, Teo KT, Yusuf S, Mann JF. The effect of ramipril and telmisartan on serum potassium and its association with cardiovascular and renal events: results from the ONTARGET trial. Eur J Prev Cardiol. 2014 Mar;21(3):299-309. doi: 10.1177/2047487313510678. Epub 2013 Nov 4. PMID 24191305
- [Derived] Dunkler D, Dehghan M, Teo KK, Heinze G, Gao P, Kohl M, Clase CM, Mann JF, Yusuf S, Oberbauer R; ONTARGET Investigators. Diet and kidney disease in high-risk individuals with type 2 diabetes mellitus. JAMA Intern Med. 2013 Oct 14;173(18):1682-92. doi: 10.1001/jamainternmed.2013.9051. PMID 23939297
- [Derived] Bohm M, Schumacher H, Laufs U, Sleight P, Schmieder R, Unger T, Teo K, Yusuf S. Effects of nonpersistence with medication on outcomes in high-risk patients with cardiovascular disease. Am Heart J. 2013 Aug;166(2):306-314.e7. doi: 10.1016/j.ahj.2013.04.016. Epub 2013 Jun 24. PMID 23895814
- [Derived] Dehghan M, Mente A, Teo KK, Gao P, Sleight P, Dagenais G, Avezum A, Probstfield JL, Dans T, Yusuf S; Ongoing Telmisartan Alone and in Combination With Ramipril Global End Point Trial (ONTARGET)/Telmisartan Randomized Assessment Study in ACEI Intolerant Subjects With Cardiovascular Disease (TRANSCEND) Trial Investigators. Relationship between healthy diet and risk of cardiovascular disease among patients on drug therapies for secondary prevention: a prospective cohort study of 31 546 high-risk individuals from 40 countries. Circulation. 2012 Dec 4;126(23):2705-12. doi: 10.1161/CIRCULATIONAHA.112.103234. PMID 23212996
- [Derived] Barzilay JI, Gao P, Clase CM, Mente A, Mann JF, Sleight P, Yusuf S, Teo KK; OnTARGET/TRANSCEND Investigators. Albuminuria and rapid loss of GFR and risk of new hip and pelvic fractures. Clin J Am Soc Nephrol. 2013 Feb;8(2):233-40. doi: 10.2215/CJN.06640712. Epub 2012 Nov 26. PMID 23184565
- [Derived] Kappert K, Bohm M, Schmieder R, Schumacher H, Teo K, Yusuf S, Sleight P, Unger T; ONTARGET/TRANSCEND Investigators. Impact of sex on cardiovascular outcome in patients at high cardiovascular risk: analysis of the Telmisartan Randomized Assessment Study in ACE-Intolerant Subjects With Cardiovascular Disease (TRANSCEND) and the Ongoing Telmisartan Alone and in Combination With Ramipril Global End Point Trial (ONTARGET). Circulation. 2012 Aug 21;126(8):934-41. doi: 10.1161/CIRCULATIONAHA.111.086660. Epub 2012 Jul 24. PMID 22829023
- [Derived] Neumann I, Grassi B. [Critically appraised article]. Rev Med Chil. 2012 Jan;140(1):117-20. Epub 2012 Apr 12. Spanish. PMID 22552566
- [Derived] Verdecchia P, Dagenais G, Healey J, Gao P, Dans AL, Chazova I, Binbrek AS, Iacobellis G, Ferreira R, Holwerda N, Karatzas N, Keltai M, Mancia G, Sleight P, Teo K, Yusuf S; Ongoing Telmisartan Alone and in Combination With Ramipril Global Endpoint TrialTelmisartan Randomized AssessmeNt Study in ACE iNtolerant subjects with cardiovascular Disease Investigators. Blood pressure and other determinants of new-onset atrial fibrillation in patients at high cardiovascular risk in the Ongoing Telmisartan Alone and in Combination With Ramipril Global Endpoint Trial/Telmisartan Randomized AssessmeNt Study in ACE iNtolerant subjects with cardiovascular Disease studies. J Hypertens. 2012 May;30(5):1004-14. doi: 10.1097/HJH.0b013e3283522a51. PMID 22495138
- [Derived] Redon J, Mancia G, Sleight P, Schumacher H, Gao P, Pogue J, Fagard R, Verdecchia P, Weber M, Bohm M, Williams B, Yusoff K, Teo K, Yusuf S; ONTARGET Investigators. Safety and efficacy of low blood pressures among patients with diabetes: subgroup analyses from the ONTARGET (ONgoing Telmisartan Alone and in combination with Ramipril Global Endpoint Trial). J Am Coll Cardiol. 2012 Jan 3;59(1):74-83. doi: 10.1016/j.jacc.2011.09.040. PMID 22192672
- [Derived] Mancia G, Schumacher H, Redon J, Verdecchia P, Schmieder R, Jennings G, Yusoff K, Ryden L, Liu GL, Teo K, Sleight P, Yusuf S. Blood pressure targets recommended by guidelines and incidence of cardiovascular and renal events in the Ongoing Telmisartan Alone and in Combination With Ramipril Global Endpoint Trial (ONTARGET). Circulation. 2011 Oct 18;124(16):1727-36. doi: 10.1161/CIRCULATIONAHA.110.008870. Epub 2011 Sep 26. PMID 21947289
- [Derived] Barzilay JI, Gao P, Ryden L, Schumacher H, Probstfield J, Commerford P, Dans A, Ferreira R, Keltai M, Paolasso E, Yusuf S, Teo K; TRANSCEND Investigators. Effects of telmisartan on glucose levels in people at high risk for cardiovascular disease but free from diabetes: the TRANSCEND study. Diabetes Care. 2011 Sep;34(9):1902-7. doi: 10.2337/dc11-0545. Epub 2011 Jul 25. PMID 21788624
- [Derived] Tobe SW, Clase CM, Gao P, McQueen M, Grosshennig A, Wang X, Teo KK, Yusuf S, Mann JF; ONTARGET and TRANSCEND Investigators. Cardiovascular and renal outcomes with telmisartan, ramipril, or both in people at high renal risk: results from the ONTARGET and TRANSCEND studies. Circulation. 2011 Mar 15;123(10):1098-107. doi: 10.1161/CIRCULATIONAHA.110.964171. Epub 2011 Feb 28. PMID 21357827
- [Derived] Barzilay JI, Gao P, O'Donnell M, Mann JF, Anderson C, Fagard R, Probstfield J, Dagenais GR, Teo K, Yusuf S; ONTARGET and TRANSCEND Investigators. Albuminuria and decline in cognitive function: The ONTARGET/TRANSCEND studies. Arch Intern Med. 2011 Jan 24;171(2):142-50. doi: 10.1001/archinternmed.2010.502. PMID 21263104
- [Derived] Dans AL, Teo K, Gao P, Chen JH, Jae-Hyung K, Yusoff K, Chaithiraphan S, Zhu J, Lisheng L, Yusuf S; Ongoing Telmisartan Alone and in Combination with Ramipril Global Endpoint Trial Investigators. In a subgroup of high-risk Asians, telmisartan was non-inferior to ramipril and better tolerated in the prevention of cardiovascular events. PLoS One. 2010 Dec 21;5(12):e13694. doi: 10.1371/journal.pone.0013694. PMID 21200437
- [Derived] Anderson C, Teo K, Gao P, Arima H, Dans A, Unger T, Commerford P, Dyal L, Schumacher H, Pogue J, Paolasso E, Holwerda N, Chazova I, Binbrek A, Young J, Yusuf S; ONTARGET and TRANSCEND Investigators. Renin-angiotensin system blockade and cognitive function in patients at high risk of cardiovascular disease: analysis of data from the ONTARGET and TRANSCEND studies. Lancet Neurol. 2011 Jan;10(1):43-53. doi: 10.1016/S1474-4422(10)70250-7. Epub 2010 Oct 25. PMID 20980201
- [Derived] Bohm M, Baumhakel M, Teo K, Sleight P, Probstfield J, Gao P, Mann JF, Diaz R, Dagenais GR, Jennings GL, Liu L, Jansky P, Yusuf S; ONTARGET/TRANSCEND Erectile Dysfunction Substudy Investigators. Erectile dysfunction predicts cardiovascular events in high-risk patients receiving telmisartan, ramipril, or both: The ONgoing Telmisartan Alone and in combination with Ramipril Global Endpoint Trial/Telmisartan Randomized AssessmeNt Study in ACE iNtolerant subjects with cardiovascular Disease (ONTARGET/TRANSCEND) Trials. Circulation. 2010 Mar 30;121(12):1439-46. doi: 10.1161/CIRCULATIONAHA.109.864199. Epub 2010 Mar 15. PMID 20231536
- [Derived] Verdecchia P, Sleight P, Mancia G, Fagard R, Trimarco B, Schmieder RE, Kim JH, Jennings G, Jansky P, Chen JH, Liu L, Gao P, Probstfield J, Teo K, Yusuf S; ONTARGET/TRANSCEND Investigators. Effects of telmisartan, ramipril, and their combination on left ventricular hypertrophy in individuals at high vascular risk in the Ongoing Telmisartan Alone and in Combination With Ramipril Global End Point Trial and the Telmisartan Randomized Assessment Study in ACE Intolerant Subjects With Cardiovascular Disease. Circulation. 2009 Oct 6;120(14):1380-9. doi: 10.1161/CIRCULATIONAHA.109.865774. Epub 2009 Sep 21. PMID 19770395
- [Derived] Sleight P, Redon J, Verdecchia P, Mancia G, Gao P, Fagard R, Schumacher H, Weber M, Bohm M, Williams B, Pogue J, Koon T, Yusuf S; ONTARGET investigators. Prognostic value of blood pressure in patients with high vascular risk in the Ongoing Telmisartan Alone and in combination with Ramipril Global Endpoint Trial study. J Hypertens. 2009 Jul;27(7):1360-9. doi: 10.1097/HJH.0b013e32832d7370. PMID 19506526
- [Derived] Mann JF, Schmieder RE, Dyal L, McQueen MJ, Schumacher H, Pogue J, Wang X, Probstfield JL, Avezum A, Cardona-Munoz E, Dagenais GR, Diaz R, Fodor G, Maillon JM, Ryden L, Yu CM, Teo KK, Yusuf S; TRANSCEND (Telmisartan Randomised Assessment Study in ACE Intolerant Subjects with Cardiovascular Disease) Investigators. Effect of telmisartan on renal outcomes: a randomized trial. Ann Intern Med. 2009 Jul 7;151(1):1-10, W1-2. doi: 10.7326/0003-4819-151-1-200907070-00122. Epub 2009 May 18. PMID 19451556
- [Derived] Telmisartan Randomised AssessmeNt Study in ACE iNtolerant subjects with cardiovascular Disease (TRANSCEND) Investigators; Yusuf S, Teo K, Anderson C, Pogue J, Dyal L, Copland I, Schumacher H, Dagenais G, Sleight P. Effects of the angiotensin-receptor blocker telmisartan on cardiovascular events in high-risk patients intolerant to angiotensin-converting enzyme inhibitors: a randomised controlled trial. Lancet. 2008 Sep 27;372(9644):1174-83. doi: 10.1016/S0140-6736(08)61242-8. Epub 2008 Aug 29. PMID 18757085
- [Derived] Mann JF, Schmieder RE, McQueen M, Dyal L, Schumacher H, Pogue J, Wang X, Maggioni A, Budaj A, Chaithiraphan S, Dickstein K, Keltai M, Metsarinne K, Oto A, Parkhomenko A, Piegas LS, Svendsen TL, Teo KK, Yusuf S; ONTARGET investigators. Renal outcomes with telmisartan, ramipril, or both, in people at high vascular risk (the ONTARGET study): a multicentre, randomised, double-blind, controlled trial. Lancet. 2008 Aug 16;372(9638):547-53. doi: 10.1016/S0140-6736(08)61236-2. PMID 18707986
- [Derived] ONTARGET Investigators; Yusuf S, Teo KK, Pogue J, Dyal L, Copland I, Schumacher H, Dagenais G, Sleight P, Anderson C. Telmisartan, ramipril, or both in patients at high risk for vascular events. N Engl J Med. 2008 Apr 10;358(15):1547-59. doi: 10.1056/NEJMoa0801317. Epub 2008 Mar 31. PMID 18378520
- [Derived] Held C, Gerstein HC, Yusuf S, Zhao F, Hilbrich L, Anderson C, Sleight P, Teo K; ONTARGET/TRANSCEND Investigators. Glucose levels predict hospitalization for congestive heart failure in patients at high cardiovascular risk. Circulation. 2007 Mar 20;115(11):1371-5. doi: 10.1161/CIRCULATIONAHA.106.661405. Epub 2007 Mar 5. PMID 17339550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the randomization visit, patients who have adhered to the medication regimen (consumed > 75% of ramipril + telmisartan during run-in phase) and were Angiotensin Converting Enzyme (ACE) tolerant were randomized into the main study (ONTARGET). ACE intolerant patients were randomized into the parallel trial (TRANSCEND).
Groups:
- Telmisartan/Ramipril (ONTARGET): Telmisartan 80mg tablet / Ramipril 10mg tablet. One tablet of each administered once daily in the morning.
- Telmisartan (ONTARGET): Telmisartan 80mg tablet /Ramipril 10mg placebo tablet. One tablet of each administered once daily in the morning.
- Ramipril (ONTARGET): Ramipril 10mg tablet / Telmisartan 80mg placebo tablet. One tablet of each administered once daily in the morning.
- Telmisartan (TRANSCEND): Telmisartan 80mg tablet, one tablet administered once daily in the morning.
- Placebo (TRANSCEND): Telmisartan 80mg placebo tablet, one tablet administered once daily in the morning.
Period: Overall Study
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET) | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Started | 8502 | 8542 | 8576 | 2954 | 2972
Completed | 8485 | 8524 | 8561 | 2946 | 2962
Not Completed | 17 | 18 | 15 | 8 | 10
Not completed — Lost to Follow-up | 14 | 14 | 12 | 5 | 5
Not completed — Withdrawal by Subject | 3 | 4 | 3 | 3 | 5

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) followed the intent-to-treat principle; it included all patients who were randomised and had any follow-up information available (i.e. 'date last seen' was available for these patients).
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET) | Telmisartan (TRANSCEND) | Placebo (TRANSCEND) | Total
Number analyzed (Participants) | 8502 | 8542 | 8576 | 2954 | 2972 | 31546
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (7.3) | 66.4 (7.1) | 66.4 (7.2) | 66.9 (7.3) | 66.9 (7.4) | 66.5 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2250 | 2250 | 2331 | 1280 | 1267 | 9378
  Male | 6252 | 6292 | 6245 | 1674 | 1705 | 22168

OUTCOME MEASURES:

1. Primary Outcome: ONTARGET. Composite Endpoint of Cardiovascular Death, Non-fatal Myocardial Infarction, Non-fatal Stroke and Hospitalization for Congestive Heart Failure
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to first event analysis of the following defined endpoints, Cardiovascular Death, Non-fatal myocardial infarction, non-fatal stroke and hospitalization for congestive heart failure.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Groups:
- Telmisartan (ONTARGET): Telmisartan 80mg tablet / Ramipril 10mg placebo tablet. One tablet of each administered once daily in the morning.
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 1386 | 1423 | 1412
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.8462, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI [0.92 to 1.07]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Non-Inferiority or Equivalence — Non-inferiority margin was 1.13; p = 0.0019, Regression, Cox; Hazard Ratio (HR) = 1.01, 97.5% CI [0.93 to 1.10]

2. Secondary Outcome: ONTARGET. Composite Endpoint of Cardiovascular Death, Non-fatal Myocardial Infarction and Non-fatal Stroke
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to first event analysis of the following defined endpoints, non-fatal myocardial infarction or non-fatal stroke
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 1200 | 1190 | 1210
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.9086, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI [0.93 to 1.09]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Non-Inferiority or Equivalence — Non-inferiority margin was 1.13; p = 0.0004, Regression, Cox; Hazard Ratio (HR) = 0.99, 97.5% CI [0.90 to 1.08]

3. Secondary Outcome: ONTARGET. Cardiovascular Death
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to the first event analysis of the endpoint cardiovascular death.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Groups:
- Telmisartan/Ramipril (ONTARGET): Telmisartan 80mg tablet /Ramipril 10mg tablet. One tablet of each administered once daily in the morning.
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 620 | 598 | 603
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.4535, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI [0.93 to 1.17]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.9421, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI [0.89 to 1.12]

4. Secondary Outcome: ONTARGET. Non-fatal Myocardial Infarction
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to the first event analysis of the endpoint non-fatal myocardial infarction.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 424 | 431 | 400
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.2909, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI [0.94 to 1.23]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.2534, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI [0.94 to 1.24]

5. Secondary Outcome: ONTARGET. Non-fatal Stroke
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to first event analysis of the endpoint non-fatal stroke.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 364 | 364 | 402
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.2248, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI [0.79 to 1.06]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.1829, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI [0.79 to 1.05]

6. Secondary Outcome: ONTARGET. Hospitalization for Congestive Heart Failure
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to the first event analysis of the endpoint hospitalization for congestive heart failure.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 332 | 394 | 354
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.4984, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI [0.82 to 1.10]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.1203, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI [0.97 to 1.29]

7. Secondary Outcome: ONTARGET. Doubling of Serum Creatinine in Diabetic Nephropathy Patients
Description: Diabetic nephropathy patients are diabetic patients with macro-albuminuria assessed as a Urinary Albumin Creatinine Ratio (UACR) ≥300 mg/g Crea at baseline.
Time Frame: 56 months
Population: FAS [DN] of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 248 | 288 | 238
participants | 30 | 24 | 23
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.4221, Regression, Cox; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.73 to 2.15]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.7305, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI [0.51 to 1.60]

8. Secondary Outcome: ONTARGET. Progression to End Stage Renal Disease (ESRD) in Diabetic Nephropathy Patients
Description: ESRD is defined by initiation of dialysis, need for renal transplantation, or eGFR <15 mL/min/1.73 m². Diabetic nephropathy patients are diabetic patients with macro-albuminuria assessed as a Urinary Albumin Creatinine Ratio (UACR) ≥300 mg/g Crea at baseline.
Time Frame: 56 months
Population: FAS [DN] of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 248 | 288 | 238
participants | 30 | 24 | 32
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.6248, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI [0.54 to 1.45]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.0751, Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.36 to 1.05]

9. Secondary Outcome: ONTARGET. All-cause Mortality in Diabetic Nephropathy Patients
Description: as for outcome 7
Time Frame: 56 months
Population: FAS [DN] of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 248 | 288 | 238
participants | 75 | 92 | 83
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.3682, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI [0.63 to 1.18]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.6014, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI [0.69 to 1.24]

10. Secondary Outcome: ONTARGET. Doubling of Serum Creatinine
Description: ONTARGET. Nephropathy subcategory: doubling of serum creatinine
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8483 | 8525 | 8557
participants | 167 | 160 | 149
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.2550, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI [0.91 to 1.42]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.5297, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI [0.86 to 1.34]

11. Secondary Outcome: ONTARGET. Progression to ESRD
Description: ONTARGET. Nephropathy subcategory: Progression to ESRD. Progression to ESRD is defined as initiation of dialysis, need for renal transplantation, or eGFR <15 mL/min/1.73 m².
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 79 | 67 | 71
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.4593, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI [0.82 to 1.56]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.7468, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI [0.68 to 1.32]

12. Primary Outcome: ONTARGET. 3-fold Composite Endpoint of Doubling of Serum Creatinine, Progression to End Stage Renal Disease (ESRD) and All-cause Mortality in Diabetic Nephropathy Patients
Description: ESRD is defined by initiation of dialysis, need for renal transplantation, or eGFR <15 mL/min/1.73 m². Diabetic nephropathy patients are diabetic patients with macro-albuminuria assessed as a Urinary Albumin Creatinine Ratio (UACR) ≥300 mg/g Crea at baseline.
  These renal outcomes were not adjudicated (apart from death).
Time Frame: 56 months
Population: Subset of the Full Analysis Set (FAS [DN]) consisting of all randomised patients with diabetic nephropathy (UACR ≥300 mg/g Crea) of the ONTARGET trial.
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 248 | 288 | 238
participants | 108 | 119 | 112
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.5461, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.71 to 1.20]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.3436, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI [0.68 to 1.14]

13. Secondary Outcome: ONTARGET. New Microalbuminuria
Description: ONTARGET. Nephropathy subcategory: New microalbuminuria. New microalbuminuria is defined as Urinary Albumin Creatinine Ratio ≥30 mg/g Crea in patients with a Urinary Albumin Creatinine Ratio <30 mg/g Crea at baseline.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 6446 | 6456 | 6532
participants | 763 | 799 | 869
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.0133, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI [0.80 to 0.97]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.1251, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI [0.84 to 1.02]

14. Secondary Outcome: ONTARGET. New Macroalbuminuria
Description: ONTARGET. Nephropathy subcategory: New macroalbuminuria. New macroalbuminuria is defined as Urinary Albumin Creatinine Ratio ≥300 mg/g Crea in patients with a Urinary Albumin Creatinine Ratio <300 mg/g Crea at baseline.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 7486 | 7465 | 7552
participants | 205 | 229 | 257
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.0213, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI [0.67 to 0.97]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.2396, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI [0.75 to 1.07]

15. Secondary Outcome: ONTARGET. Combined Endpoint of Doubling of Serum Creatinine, Progression to ESRD, New Microalbuminuria, or New Macroalbuminuria
Description: ONTARGET. Nephropathy subcategory: Combined endpoint of doubling of serum creatinine, progression to ESRD, new microalbuminuria, or new macroalbuminuria
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 1067 | 1101 | 1190
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.0111, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI [0.83 to 0.98]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.0606, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI [0.85 to 1.00]

16. Secondary Outcome: ONTARGET. Normalisation From Micro- or Macroalbuminuria to Normoalbuminuria
Description: ONTARGET. Nephropathy subcategory: Normalisation from micro- or macroalbuminuria to normoalbuminuria. Normalisation from micro- or macroalbuminuria to normoalbuminuria is defined as UACR <30 mg/g Crea in patients with a UACR ≥30 mg/g Crea at baseline.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 1337 | 1361 | 1314
participants | 508 | 483 | 448
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.0082, Regression, Cox; Hazard Ratio (HR) = 1.19, 95% CI [1.05 to 1.35]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.2164, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI [0.95 to 1.23]

17. Secondary Outcome: ONTARGET. Newly Diagnosed Congestive Heart Failure
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to the first event analysis of the endpoint Newly diagnosed Congestive Heart failure.
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 469 | 529 | 503
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.3732, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI [0.83 to 1.07]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.3633, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI [0.94 to 1.20]

18. Secondary Outcome: ONTARGET. Cardiovascular Revascularization Procedure
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET).
Time Frame: 56 months
Population: FAS of the ONTARGET trial
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8502 | 8542 | 8576
participants | 1303 | 1290 | 1269
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.2713, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI [0.97 to 1.13]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); Test type: Superiority or Other; p = 0.5150, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI [0.95 to 1.11]

19. Secondary Outcome: ONTARGET. Newly Diagnosed Diabetes
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to the first event analysis of the endpoint Newly diagnosed Diabetes. Only calculated for those patients without diabetes at baseline.
Time Frame: 56 months
Population: Only patients of the ONTARGET trial treated with Telmisartan 80mg/ramipril 10mg or Telmisartan 80mg/Ramipril 10mg placebo or Ramipril 10mg/ telmisartan 80mg placebo daily for 56 months without baseline diabetes.
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 5037 | 4992 | 5123
participants | 224 | 277 | 249
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); for subjects without diabetes at baseline; Test type: Superiority or Other; p = 0.3485, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI [0.77 to 1.10]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); for subjects without diabetes at baseline; Test type: Superiority or Other; p = 0.1235, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI [0.96 to 1.36]

20. Secondary Outcome: ONTARGET. Cognitive Decline
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to first event analysis of the endpoint cognitive decline i.e. Comparison of the Mini mental state Evaluation (MMSE) of patients at baseline with that at the 2years and end of trial. A decrease in MMSE from baseline represents a cognitive decline. This outcome measure is only available for those patients who had MMSE at baseline.
Time Frame: 56 months
Population: Only patients of the ONTARGET trial treated with Telmisartan 80mg/ramipril 10mg or Telmisartan 80mg/Ramipril 10mg placebo or Ramipril 10mg/ telmisartan 80mg placebo daily for 56 months with Mini mental state evaluation (MMSE) at baseline.
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 7461 | 7566 | 7602
participants | 561 | 600 | 577
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); for subjects with available Mini Mental State Examination (MMSE) at baseline; Test type: Superiority or Other; p = 0.8690, Chi-squared; Risk Ratio (RR) = 0.99, 95% CI [0.89 to 1.11]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); for subjects with available Mini Mental State Examination (MMSE) at baseline; Test type: Superiority or Other; p = 0.4337, Chi-squared; Risk Ratio (RR) = 1.04, 95% CI [0.94 to 1.17]

21. Secondary Outcome: ONTARGET. New Onset of Atrial Fibrillation
Description: The Ongoing Telmisartan Alone and combination with Ramipril global Endpoint trial (ONTARGET). Time to first event analysis of endpoint new onset of atrial fibrillation.
Time Frame: 56 months
Population: Only patients of the ONTARGET trial treated with Telmisartan 80mg/ramipril 10mg or Telmisartan 80mg/Ramipril 10mg placebo or Ramipril 10mg/ telmisartan 80mg placebo daily for 56 months without atrial fibrillation at baseline.
Measure: Number; unit: participants
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET)
Number analyzed (Participants) | 8218 | 8259 | 8296
participants | 542 | 560 | 586
Statistical Analysis 1: Comparison: Telmisartan/Ramipril (ONTARGET) vs Ramipril (ONTARGET); for subjects without atrial fibrillation at baseline; Test type: Superiority or Other; p = 0.2666, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI [0.83 to 1.05]
Statistical Analysis 2: Comparison: Telmisartan (ONTARGET) vs Ramipril (ONTARGET); for subjects without atrial fibrillation at baseline; Test type: Superiority or Other; p = 0.4784, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI [0.85 to 1.08]

22. Secondary Outcome: TRANSCEND. Composite Endpoint of Cardiovascular Death, Non-fatal Myocardial Infarction and Non-fatal Stroke
Description: Telmisartan Randomized Assessment Study in Angiotension Converting Enzyme inhibitor intolerant subjects with cardiovascular disease (TRANSCEND). Time to first event analysis of the following defined endpoints, Cardiovascular Death, Non-fatal myocardial infarction, non-fatal stroke and hospitalization for congestive heart failure.
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 384 | 440
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0483, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI [0.76 to 1.00]

23. Primary Outcome: TRANSCEND. Composite Endpoint of Cardiovascular Death, Non-fatal Myocardial Infarction, Non-fatal Stroke and Hospitalization for Congestive Heart Failure
Description: as for outcome 22
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 465 | 504
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.2192, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI [0.81 to 1.05]

24. Secondary Outcome: TRANSCEND. Cardiovascular Death
Description: Telmisartan Randomized Assessment Study in Angiotension Converting Enzyme inhibitor intolerant subjects with cardiovascular disease (TRANSCEND). Time to the first event analysis of the endpoint cardiovascular death.
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 227 | 223
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.7764, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI [0.85 to 1.24]

25. Secondary Outcome: TRANSCEND. Non-fatal Myocardial Infarction
Description: Telmisartan Randomized Assessment Study in Angiotension Converting Enzyme inhibitor intolerant subjects with cardiovascular disease (TRANSCEND). Time to the first event analysis of the endpoint non-fatal myocardial infarction.
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 114 | 145
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0574, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI [0.62 to 1.01]

26. Secondary Outcome: TRANSCEND. Non-fatal Stroke
Description: Telmisartan Randomized Assessment Study in Angiotension Converting Enzyme inhibitor intolerant subjects with cardiovascular disease (TRANSCEND).
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 112 | 136
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.1365, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI [0.64 to 1.06]

27. Secondary Outcome: TRANSCEND. Hospitalization for Congestive Heart Failure
Description: as for outcome 26
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 134 | 129
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.6940, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI [0.82 to 1.34]

28. Secondary Outcome: TRANSCEND. Doubling of Serum Creatinine
Description: TRANSCEND. Nephropathy subcategory: doubling of serum creatinine
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2950 | 2965
participants | 62 | 40
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0245, Regression, Cox; Hazard Ratio (HR) = 1.58, 95% CI [1.06 to 2.35]

29. Secondary Outcome: TRANSCEND. Progression to ESRD
Description: TRANSCEND. Nephropathy subcategory: Progression to ESRD. Progression to ESRD is defined as initiation of dialysis, need for renal transplantation, or eGFR <15 mL/min/1.73m²
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 11 | 14
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.5798, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI [0.36 to 1.76]

30. Secondary Outcome: TRANSCEND. New Microalbuminuria
Description: TRANSCEND. Nephropathy subcategory: New microalbuminuria. New microalbuminuria is defined as UACR ≥30 mg/g creatinine [Crea] in patients with a UACR <30 mg/g Crea at baseline
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2372 | 2403
participants | 276 | 363
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0006, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI [0.65 to 0.89]

31. Secondary Outcome: TRANSCEND. New Macroalbuminuria
Description: TRANSCEND. Nephropathy subcategory: New macroalbuminuria. New macroalbuminuria is defined as UACR ≥300 mg/g creatinine [Crea] in patients with a UACR <300 mg/g Crea at baseline
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2658 | 2676
participants | 66 | 101
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0085, Regression, Cox; Hazard Ratio (HR) = 0.66, 95% CI [0.48 to 0.90]

32. Secondary Outcome: TRANSCEND. Combined Endpoint of Doubling Serum Creatinine, Progression to ESRD, New Microalbuminuria or New Macroalbuminuria
Description: TRANSCEND. Nephropathy subcategory: Combined endpoint of doubling serum creatinine, progression to ESRD, new microalbuminuria or new macroalbuminuria
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 357 | 448
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0015, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI [0.69 to 0.92]

33. Secondary Outcome: TRANSCEND. Normalisation From Micro- or Macroalbuminuria to Normoalbuminuria
Description: TRANSCEND. Nephropathy subcategory: Normalisation from micro- or macroalbuminuria to normoalbuminuria. Normalisation from micro- or macroalbuminuria to normoalbuminuria is defined as UACR <30 mg/g Crea in patients with a UACR ≥30 mg/g Crea at baseline.
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 319 | 318
participants | 135 | 110
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0101, Regression, Cox; Hazard Ratio (HR) = 1.39, 95% CI [1.08 to 1.79]

34. Secondary Outcome: TRANSCEND. New Onset of Atrial Fibrillation
Description: as for outcome 26
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2851 | 2870
participants | 181 | 182
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.9563, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI [0.82 to 1.24]

35. Secondary Outcome: TRANSCEND. Cognitive Decline
Description: Telmisartan Randomized Assessment Study in Angiotension Converting Enzyme inhibitor intolerant subjects with cardiovascular disease (TRANSCEND). Time to first event analysis of the endpoint cognitive decline i.e. Comparison of the Mini mental state Evaluation (MMSE) of patients at baseline with that at the 2years and end of trial. A decrease in MMSE from baseline represents a cognitive decline. This outcome measure is only available for those patients who had MMSE at baseline.
Time Frame: 56 months
Population: Only patients of the TRANSCEND trial treated with Telmisartan 80mg or telmisartan 80mg placebo daily for 56 months with Mini mental state evaluation (MMSE) at baseline.
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2642 | 2589
participants | 230 | 192
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0868, Chi-squared; Risk Ratio (RR) = 1.17, 95% CI [0.98 to 1.41]

36. Secondary Outcome: TRANSCEND. Newly Diagnosed Diabetes
Description: Telmisartan Randomized Assessment Study in Angiotension Converting Enzyme inhibitor intolerant subjects with cardiovascular disease (TRANSCEND). Time to the first event analysis of the endpoint Newly diagnosed Diabetes. Only calculated for those patients without diabetes at baseline.
Time Frame: 56 months
Population: Only for patients of TRANSCEND trial treated with Telmisartan 80mg or Telmisartan 80mg placebo daily for 56 months without diabetes at baseline.
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 1710 | 1751
participants | 124 | 165
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.0172, Regression, Cox; Hazard Ratio (HR) = 0.75, 95% CI [0.60 to 0.95]

37. Secondary Outcome: TRANSCEND. Cardiovascular Revascularization Procedure
Description: as for outcome 26
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2954 | 2972
participants | 351 | 390
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.1431, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI [0.78 to 1.04]

38. Secondary Outcome: TRANSCEND. Newly Diagnosed Congestive Heart Failure
Description: as for outcome 26
Time Frame: 56 months
Population: FAS of the TRANSCEND trial
Measure: Number; unit: participants
Arm/Group | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Number analyzed (Participants) | 2949 | 2965
participants | 187 | 191
Statistical Analysis 1: Comparison: Telmisartan (TRANSCEND) vs Placebo (TRANSCEND); Test type: Superiority or Other; p = 0.8974, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI [0.81 to 1.21]

ADVERSE EVENTS:
Time Frame: Up to 6 Years
Description: In the ONTARGET part, the time frame is up to 5.5 years and in the TRANSCEND part up to 6 years
Arm/Group | Telmisartan/Ramipril (ONTARGET) | Telmisartan (ONTARGET) | Ramipril (ONTARGET) | Telmisartan (TRANSCEND) | Placebo (TRANSCEND)
Serious Adverse Events (participants affected / at risk) | 5268/8502 | 5506/8542 | 5375/8576 | 1781/2954 | 1830/2972
Other Adverse Events (participants affected / at risk) | 0/8502 | 0/8542 | 0/8576 | 0/2954 | 0/2972
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan/Ramipril (ONTARGET) (N=8502) | Telmisartan (ONTARGET) (N=8542) | Ramipril (ONTARGET) (N=8576) | Telmisartan (TRANSCEND) (N=2954) | Placebo (TRANSCEND) (N=2972)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 125 | 156 | 131 | 43 | 36
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0 | 0
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hyperglobulinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hypersplenism (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 6 | 8 | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 4 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 3 | 1 | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 4 | 3 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 8 | 1 | 2 | 1 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Red blood cell abnormality (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Spleen disorder (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4 | 3 | 3 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 1
AV dissociation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 6 | 11 | 7 | 1 | 3
Acute left ventricular failure (Cardiac disorders) | 0 | 4 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 1 | 0 | 1
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1206 | 1296 | 1244 | 418 | 455
Angina unstable (Cardiac disorders) | 7 | 15 | 12 | 0 | 5
Aortic valve disease (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 2 | 5 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 3 | 7 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 38 | 41 | 41 | 19 | 15
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 2 | 2 | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 449 | 499 | 509 | 146 | 149
Atrial flutter (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 6 | 4 | 7 | 3 | 2
Atrioventricular block complete (Cardiac disorders) | 18 | 18 | 11 | 3 | 2
Atrioventricular block first degree (Cardiac disorders) | 3 | 0 | 2 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 4 | 6 | 4 | 1 | 2
Bifascicular block (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Bradyarrhythmia (Cardiac disorders) | 5 | 2 | 2 | 2 | 1
Bradycardia (Cardiac disorders) | 30 | 30 | 32 | 8 | 10
Bundle branch block bilateral (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac aneurysm (Cardiac disorders) | 2 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 35 | 37 | 37 | 12 | 9
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 11 | 6 | 7 | 2 | 5
Cardiac failure acute (Cardiac disorders) | 47 | 27 | 52 | 26 | 15
Cardiac failure chronic (Cardiac disorders) | 0 | 2 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 400 | 484 | 465 | 174 | 172
Cardiac pseudoaneurysm (Cardiac disorders) | 0 | 2 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 4 | 0 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac valve sclerosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 8 | 7 | 2 | 1 | 3
Cardiogenic shock (Cardiac disorders) | 7 | 6 | 9 | 2 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 2 | 2 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 1 | 1 | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery dilatation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 12 | 15 | 9 | 5 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Diabetic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 3 | 2 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 0 | 2 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 4 | 1 | 0 | 2
Left ventricular failure (Cardiac disorders) | 0 | 1 | 3 | 0 | 3
Low cardiac output syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 3 | 1 | 2 | 0 | 2
Myocardial infarction (Cardiac disorders) | 456 | 480 | 457 | 138 | 161
Myocardial ischaemia (Cardiac disorders) | 11 | 9 | 11 | 4 | 4
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 3 | 0 | 0 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pacemaker generated arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 7 | 13 | 5 | 2 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2 | 3 | 1 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 1 | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 4 | 4 | 3 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 11 | 9 | 12 | 4 | 1
Sinus arrest (Cardiac disorders) | 1 | 2 | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 2 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 6 | 6 | 5 | 5 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 2 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 2 | 0 | 1
Tachycardia (Cardiac disorders) | 6 | 1 | 3 | 0 | 0
Trifascicular block (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 62 | 75 | 64 | 18 | 24
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 3 | 1 | 0 | 1 | 0
Ventricular remodeling (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 19 | 19 | 15 | 6 | 1
Ventricular tachycardia (Cardiac disorders) | 7 | 5 | 2 | 0 | 1
Wandering pacemaker (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Alagille syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 2 | 1 | 0 | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 3 | 0 | 0 | 0 | 0
Dolichocolon (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Fragile X syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 3 | 5 | 1 | 0 | 0
Kidney malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Limb reduction defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Meningomyelocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Neural tube defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Oculopharyngeal dystrophy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Osteogenesis imperfecta (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 3 | 1 | 0 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 0 | 0
Transposition of the great vessels (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Turner's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0 | 0 | 2 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 2 | 0 | 0
Middle ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 28 | 18 | 30 | 13 | 18
Vertigo labyrinthine (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 2 | 1 | 0 | 2 | 1
Vestibular ataxia (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Vestibular neuronitis (Ear and labyrinth disorders) | 3 | 3 | 0 | 0 | 0
Addison's disease (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 1 | 1 | 0 | 0
Adrenal mass (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Antidiuretic hormone abnormality (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Endocrine disorder (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 2 | 1 | 4 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 6 | 5 | 9 | 1 | 1
Hypopituitarism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 4 | 7 | 4 | 2 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Thyroid cyst (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | 1 | 0 | 0 | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 1 | 1 | 0 | 0
Blindness (Eye disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 12 | 10 | 15 | 4 | 1
Cataract diabetic (Eye disorders) | 0 | 0 | 2 | 1 | 0
Choroidal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Corneal infiltrates (Eye disorders) | 0 | 0 | 0 | 1 | 0
Diabetic retinal oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 3 | 3 | 5 | 2 | 3
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Endocrine ophthalmopathy (Eye disorders) | 0 | 1 | 0 | 0 | 0
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye degenerative disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 3 | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 1 | 0 | 0
Glaucoma (Eye disorders) | 3 | 12 | 6 | 3 | 2
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0
Macular degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 1
Maculopathy (Eye disorders) | 1 | 1 | 0 | 0 | 0
Miosis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Open angle glaucoma (Eye disorders) | 0 | 1 | 2 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 1 | 0
Optic neuropathy (Eye disorders) | 0 | 0 | 0 | 1 | 0
Pseudophakia (Eye disorders) | 0 | 0 | 2 | 0 | 0
Pterygium (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal artery embolism (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 2 | 0 | 0
Retinal artery thrombosis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 6 | 8 | 0 | 1 | 0
Retinal disorder (Eye disorders) | 1 | 1 | 0 | 0 | 0
Retinal infarction (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal ischaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal neovascularisation (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal vascular thrombosis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0 | 1 | 0 | 0
Retinopathy (Eye disorders) | 4 | 6 | 4 | 1 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinopathy proliferative (Eye disorders) | 0 | 0 | 0 | 1 | 0
Swollen tear duct (Eye disorders) | 0 | 0 | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1 | 1 | 1 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1 | 0 | 0
Visual disturbance (Eye disorders) | 2 | 0 | 1 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 1 | 0 | 0
Vitreous opacities (Eye disorders) | 0 | 0 | 2 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 3 | 4 | 5 | 1 | 2
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 43 | 23 | 39 | 4 | 10
Abdominal pain lower (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 17 | 22 | 15 | 8 | 2
Acute abdomen (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal dilatation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Anal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis perforated (Gastrointestinal disorders) | 2 | 3 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 3 | 3 | 3 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 8 | 6 | 7 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 4 | 2 | 12 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 3 | 2 | 0 | 2 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 4 | 6 | 5 | 2 | 3
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 15 | 10 | 19 | 2 | 6
Crohn's disease (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Diabetic gastropathy (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 45 | 39 | 32 | 12 | 3
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 4 | 7 | 7 | 5 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 3 | 4 | 5 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1
Diverticulum oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 15 | 13 | 11 | 5 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 6 | 4 | 3 | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 8 | 1 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 8 | 5 | 5 | 1
Dysphagia (Gastrointestinal disorders) | 7 | 5 | 9 | 1 | 1
Enteritis (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 1
Enterocele (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enterocolonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 4 | 2 | 1 | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 5 | 8 | 5 | 2 | 3
Gastric hypermotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 24 | 26 | 23 | 6 | 5
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 5 | 10 | 8 | 7 | 3
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 25 | 31 | 28 | 7 | 15
Gastritis erosive (Gastrointestinal disorders) | 4 | 6 | 2 | 3 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 56 | 59 | 50 | 19 | 11
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 4 | 3 | 3 | 0 | 0
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastrointestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 3 | 3 | 0 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 18 | 9 | 10 | 4 | 2
Gastroptosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 8 | 8 | 8 | 2 | 2
Haematochezia (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 7 | 9 | 5 | 7 | 6
Hiatus hernia (Gastrointestinal disorders) | 8 | 6 | 3 | 3 | 3
Hiatus hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 4 | 7 | 4 | 2 | 7
Ileus paralytic (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 21 | 34 | 26 | 2 | 9
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Intestinal angina (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Intestinal functional disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 13 | 14 | 11 | 3 | 3
Intestinal perforation (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1
Jejunitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 8 | 4 | 11 | 2 | 2
Mesenteric artery embolism (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Mesenteric occlusion (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth cyst (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 19 | 24 | 20 | 6 | 7
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Oesophageal dilatation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal disorder (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Oesophageal dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Oesophageal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal rupture (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 5 | 16 | 6 | 3 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 17 | 20 | 13 | 3 | 2
Pancreatitis acute (Gastrointestinal disorders) | 8 | 11 | 7 | 4 | 5
Pancreatitis chronic (Gastrointestinal disorders) | 2 | 3 | 5 | 2 | 4
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 9 | 5 | 10 | 3 | 4
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 | 3 | 2 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Periproctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Peritoneal effusion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 4 | 2 | 5 | 2 | 2
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Proctocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 19 | 10 | 9 | 3 | 8
Rectal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 3 | 2 | 2 | 1 | 4
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 11 | 12 | 5 | 0 | 3
Small intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 4 | 1 | 2 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 4 | 7 | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 16 | 19 | 16 | 8 | 6
Uraemic gastropathy (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 27 | 28 | 29 | 6 | 6
Abasia (General disorders) | 0 | 1 | 0 | 0 | 0
Accidental death (General disorders) | 0 | 0 | 1 | 0 | 0
Adverse drug reaction (General disorders) | 2 | 1 | 1 | 0 | 0
Application site bleeding (General disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 17 | 15 | 20 | 7 | 4
Cardiac death (General disorders) | 1 | 2 | 0 | 0 | 0
Chest discomfort (General disorders) | 7 | 4 | 11 | 3 | 3
Chest pain (General disorders) | 117 | 96 | 103 | 38 | 26
Chills (General disorders) | 2 | 0 | 1 | 0 | 0
Chronic fatigue syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 31 | 32 | 31 | 11 | 8
Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Drowning (General disorders) | 1 | 1 | 0 | 1 | 1
Drug interaction (General disorders) | 0 | 3 | 0 | 0 | 0
Drug intolerance (General disorders) | 2 | 0 | 0 | 0 | 0
Electrocution (General disorders) | 0 | 0 | 2 | 0 | 0
Exercise tolerance decreased (General disorders) | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 9 | 3 | 8 | 1 | 1
Gait deviation (General disorders) | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 4 | 2 | 1 | 0 | 0
General physical health deterioration (General disorders) | 6 | 6 | 1 | 3 | 1
Generalised oedema (General disorders) | 1 | 0 | 2 | 1 | 0
Granuloma (General disorders) | 0 | 0 | 0 | 0 | 1
Hernia (General disorders) | 4 | 11 | 4 | 0 | 2
Hernia obstructive (General disorders) | 0 | 1 | 0 | 0 | 1
Hyperthermia (General disorders) | 1 | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 2 | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 2 | 1 | 0 | 0
Implant site effusion (General disorders) | 1 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic ulcer (General disorders) | 1 | 1 | 1 | 0 | 0
Loss of control of legs (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 6 | 9 | 2 | 1 | 0
Mass (General disorders) | 0 | 0 | 1 | 0 | 0
Microlithiasis (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 3 | 0 | 0 | 0
Multi-organ failure (General disorders) | 9 | 8 | 11 | 3 | 3
Necrosis (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 29 | 33 | 29 | 13 | 12
Oedema (General disorders) | 1 | 2 | 1 | 0 | 1
Oedema peripheral (General disorders) | 4 | 9 | 8 | 0 | 0
Orthostatic intolerance (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 4 | 1 | 0 | 1 | 1
Pre-existing disease (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 30 | 21 | 23 | 4 | 2
Secretion discharge (General disorders) | 0 | 1 | 0 | 0 | 0
Submandibular mass (General disorders) | 1 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 134 | 155 | 141 | 69 | 68
Sudden death (General disorders) | 11 | 14 | 12 | 2 | 3
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0 | 0
Ulcer (General disorders) | 1 | 1 | 3 | 0 | 1
Ulcer haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 2 | 3 | 0 | 0 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 2 | 5 | 1 | 3
Biliary colic (Hepatobiliary disorders) | 2 | 3 | 3 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Biliary ischaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 9 | 2 | 5 | 3 | 1
Cholangitis acute (Hepatobiliary disorders) | 2 | 1 | 2 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 20 | 26 | 41 | 12 | 9
Cholecystitis acute (Hepatobiliary disorders) | 11 | 18 | 12 | 3 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 3 | 3 | 1 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 28 | 32 | 21 | 13 | 9
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 4 | 0 | 0
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 3 | 1 | 0 | 0 | 1
Gallbladder necrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 7 | 6 | 3 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 7 | 3 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 0
Jaundice (Hepatobiliary disorders) | 3 | 5 | 5 | 2 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 4 | 1 | 2 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 2 | 1 | 0 | 3
Portal hypertension (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Portal vein phlebitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Allergic oedema (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 2 | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Anaphylactoid shock (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 3 | 1 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 2 | 4 | 1 | 1
Immunodeficiency (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Insulin autoimmune syndrome (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Pancreas transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 3 | 2 | 1 | 1 | 2
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Abscess (Infections and infestations) | 1 | 2 | 2 | 2 | 0
Abscess intestinal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 1 | 3 | 0 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Anogenital warts (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Appendiceal abscess (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 14 | 8 | 11 | 4 | 4
Application site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arteriosclerotic gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 3 | 1 | 5 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Aspergilloma (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 3 | 3 | 2 | 1 | 0
Bacterial food poisoning (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bone tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Bronchiectasis (Infections and infestations) | 2 | 1 | 2 | 2 | 0
Bronchitis (Infections and infestations) | 37 | 30 | 35 | 16 | 12
Bronchitis viral (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 26 | 25 | 21 | 6 | 8
Bursitis infective (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Campylobacter intestinal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Carbuncle (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cavernous sinus thrombosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 26 | 29 | 39 | 12 | 14
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Cellulitis orbital (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Central nervous system infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 4 | 0 | 1 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Citrobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 1 | 4 | 1 | 2
Creutzfeldt-Jakob disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 5 | 7 | 10 | 5 | 4
Dengue fever (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 2 | 2 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 18 | 16 | 22 | 5 | 6
Ear infection (Infections and infestations) | 5 | 4 | 0 | 0 | 1
Empyema (Infections and infestations) | 3 | 1 | 5 | 1 | 0
Encephalitis viral (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 3 | 0 | 2 | 2 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enterobacter pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 9 | 13 | 10 | 3 | 3
Escherichia bacteraemia (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
External ear cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Extradural abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 2 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gallbladder abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 2 | 0 | 1
Gastric infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 46 | 33 | 32 | 8 | 11
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 2 | 3 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 2 | 4 | 1 | 0 | 0
Genital infection female (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Genitourinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Graft infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Groin infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 5 | 8 | 10 | 6 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Herpes zoster infection neurological (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Histoplasmosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Incision site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Incisional hernia gangrenous (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infected lymphocele (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 10 | 18 | 23 | 2 | 3
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 2 | 2 | 0 | 1
Influenza (Infections and infestations) | 4 | 5 | 3 | 0 | 3
Injection site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Injection site infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Intestinal fistula infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Intestinal gangrene (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 2 | 3 | 2 | 3 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 2 | 1 | 0
Leptospirosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 3 | 1 | 4 | 0 | 0
Lobar pneumonia (Infections and infestations) | 9 | 11 | 14 | 2 | 5
Localised infection (Infections and infestations) | 3 | 3 | 7 | 3 | 2
Lower respiratory tract infection (Infections and infestations) | 22 | 26 | 23 | 10 | 8
Lung abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 2 | 3 | 5 | 1 | 3
Lung infection pseudomonal (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Meningoencephalitis herpetic (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Mycotic corneal ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Myringitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 6 | 2 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Neurosyphilis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nocardiosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nosocomial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 3 | 2 | 1 | 2
Osteomyelitis (Infections and infestations) | 2 | 2 | 6 | 1 | 1
Osteomyelitis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Pancreas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Perianal abscess (Infections and infestations) | 5 | 4 | 1 | 0 | 0
Peridiverticular abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Peritoneal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Peritoneal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 2 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 272 | 310 | 278 | 99 | 97
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 3 | 2 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 2 | 2 | 0 | 0
Post procedural infection (Infections and infestations) | 4 | 4 | 7 | 0 | 3
Postoperative abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Postoperative wound infection (Infections and infestations) | 4 | 7 | 12 | 2 | 2
Prostate infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Prostatic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 3 | 3 | 6 | 2 | 2
Purulence (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 15 | 15 | 10 | 8 | 6
Pyelonephritis acute (Infections and infestations) | 2 | 2 | 2 | 3 | 0
Pyelonephritis chronic (Infections and infestations) | 4 | 1 | 7 | 3 | 3
Pyothorax (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Renal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 14 | 15 | 15 | 11 | 6
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 2 | 2 | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Scrub typhus (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 49 | 43 | 32 | 14 | 9
Septic shock (Infections and infestations) | 7 | 14 | 16 | 7 | 3
Sinusitis (Infections and infestations) | 1 | 2 | 7 | 0 | 1
Skin infection (Infections and infestations) | 2 | 2 | 0 | 0 | 1
Small intestine gangrene (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 4 | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Syphilitic endocarditis of heart valve (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tick-borne fever (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Toxoplasmosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Tracheobronchitis (Infections and infestations) | 1 | 1 | 3 | 0 | 0
Tuberculosis (Infections and infestations) | 4 | 2 | 2 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 10 | 11 | 6 | 4
Urethral carbuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urethritis (Infections and infestations) | 1 | 2 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 73 | 71 | 79 | 31 | 26
Urinary tract infection enterococcal (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Urogenital infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 14 | 11 | 7 | 3 | 4
Vaginal abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 4 | 2 | 3 | 2 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Wound abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 2 | 6 | 5 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Accident at home (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Accident at work (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Accidental needle stick (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 1 | 0
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 10 | 16 | 12 | 1 | 4
Arterial injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0
Asbestosis (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 1 | 1
Blast injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 5 | 2 | 1 | 0 | 0
Burn of internal organs (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 1 | 0
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 3 | 4 | 3 | 0 | 1
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 4 | 1 | 3 | 0 | 0
Confusion postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 9 | 5 | 2 | 2
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Cranial nerve injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1
Device breakage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Device electrical finding (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Device migration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Device occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 3 | 3 | 3 | 1 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Eye penetration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 3 | 8 | 2 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 97 | 99 | 98 | 38 | 37
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 3 | 4 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 17 | 14 | 15 | 6 | 5
Fibula fracture (Injury, poisoning and procedural complications) | 5 | 4 | 2 | 4 | 1
Foot fracture (Injury, poisoning and procedural complications) | 3 | 6 | 5 | 1 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 3 | 4 | 1 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 4 | 6 | 4 | 2 | 3
Head injury (Injury, poisoning and procedural complications) | 11 | 9 | 6 | 7 | 6
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 55 | 47 | 43 | 21 | 18
Humerus fracture (Injury, poisoning and procedural complications) | 14 | 11 | 8 | 2 | 3
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 2
Injury (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 1
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 6 | 10 | 4 | 1 | 3
Joint injury (Injury, poisoning and procedural complications) | 1 | 7 | 10 | 3 | 2
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 12 | 4 | 6 | 5 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0
Lung injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 0 | 1
Mountain sickness acute (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 5 | 2 | 0 | 0
Pacemaker complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 5 | 3 | 4 | 0 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 5 | 6 | 8 | 0 | 3
Pelvic organ injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 4 | 2 | 1 | 2
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 1 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 2 | 3 | 1 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 5 | 4 | 2 | 0 | 2
Reocclusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 18 | 19 | 16 | 2 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 23 | 11 | 18 | 5 | 6
Scapula fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0
Sciatic nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Silicosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 3 | 8 | 4 | 2 | 1
Skull fracture (Injury, poisoning and procedural complications) | 5 | 3 | 5 | 3 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 19 | 17 | 23 | 5 | 4
Splenic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Spondylopathy traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 0
Sternal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 8 | 9 | 11 | 3 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 3 | 0
Tendon injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 3 | 2 | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2 | 3 | 4 | 3 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 0 | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 6 | 6 | 2 | 2 | 5
Traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Traumatic anuria (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 2 | 0 | 4 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 12 | 8 | 14 | 7 | 5
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Urinary tract injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Vertebral injury (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 1
Whiplash injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 9 | 3 | 7 | 1 | 2
Acid base balance abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Amphetamines positive (Investigations) | 0 | 0 | 1 | 0 | 0
Angiogram (Investigations) | 85 | 79 | 72 | 35 | 22
Angiogram cerebral (Investigations) | 1 | 0 | 1 | 0 | 0
Angiogram peripheral (Investigations) | 7 | 6 | 6 | 0 | 2
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 | 0 | 0 | 0
Aortogram (Investigations) | 1 | 1 | 0 | 0 | 0
Arteriogram (Investigations) | 2 | 4 | 3 | 0 | 2
Arteriogram carotid (Investigations) | 3 | 3 | 8 | 3 | 1
Arteriogram coronary (Investigations) | 64 | 68 | 55 | 18 | 26
Arteriogram coronary abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Arteriogram renal (Investigations) | 3 | 2 | 0 | 0 | 1
Arthroscopy (Investigations) | 6 | 13 | 12 | 6 | 3
Aspiration bronchial (Investigations) | 0 | 0 | 0 | 0 | 1
Barium enema (Investigations) | 0 | 0 | 1 | 0 | 0
Barium meal normal (Investigations) | 0 | 1 | 0 | 0 | 0
Biopsy (Investigations) | 4 | 4 | 3 | 0 | 0
Biopsy artery (Investigations) | 1 | 0 | 0 | 0 | 0
Biopsy bladder (Investigations) | 0 | 1 | 0 | 1 | 0
Biopsy brain (Investigations) | 0 | 1 | 1 | 0 | 0
Biopsy breast (Investigations) | 0 | 0 | 1 | 0 | 1
Biopsy cervix (Investigations) | 0 | 0 | 1 | 0 | 0
Biopsy kidney (Investigations) | 1 | 2 | 0 | 0 | 0
Biopsy larynx (Investigations) | 0 | 1 | 0 | 0 | 0
Biopsy liver (Investigations) | 0 | 0 | 3 | 0 | 1
Biopsy lung (Investigations) | 3 | 3 | 2 | 0 | 0
Biopsy lymph gland (Investigations) | 0 | 0 | 1 | 0 | 0
Biopsy muscle (Investigations) | 0 | 0 | 1 | 0 | 0
Biopsy oesophagus (Investigations) | 2 | 0 | 0 | 0 | 0
Biopsy pleura (Investigations) | 0 | 0 | 1 | 0 | 0
Biopsy prostate (Investigations) | 5 | 2 | 5 | 0 | 1
Biopsy site unspecified normal (Investigations) | 0 | 1 | 0 | 0 | 0
Biopsy spinal cord (Investigations) | 0 | 1 | 0 | 0 | 0
Biopsy tongue (Investigations) | 1 | 0 | 0 | 0 | 0
Biopsy trachea (Investigations) | 1 | 0 | 0 | 0 | 0
Biopsy uterus (Investigations) | 0 | 0 | 0 | 2 | 0
Biopsy vulva (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alcohol increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase MB normal (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 43 | 29 | 30 | 9 | 3
Blood culture positive (Investigations) | 1 | 0 | 1 | 0 | 1
Blood glucose fluctuation (Investigations) | 1 | 0 | 2 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood immunoglobulin G increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood osmolarity decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood phosphorus (Investigations) | 0 | 1 | 0 | 0 | 0
Blood potassium abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood potassium increased (Investigations) | 3 | 1 | 2 | 0 | 0
Blood pressure abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 2 | 1 | 0 | 1
Blood pressure orthostatic (Investigations) | 1 | 0 | 0 | 0 | 0
Blood pressure orthostatic abnormal (Investigations) | 0 | 0 | 2 | 0 | 0
Blood sodium abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood sodium increased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood urea (Investigations) | 0 | 1 | 0 | 0 | 0
Blood urea abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 7 | 1 | 5 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urine (Investigations) | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 1 | 0 | 0
Borrelia burgdorferi serology positive (Investigations) | 0 | 0 | 1 | 0 | 0
Bronchoscopy (Investigations) | 3 | 0 | 2 | 1 | 0
Cardiac electrophysiologic study (Investigations) | 0 | 8 | 0 | 2 | 1
Cardiac enzymes increased (Investigations) | 0 | 0 | 0 | 1 | 0
Cardiac function test (Investigations) | 0 | 1 | 0 | 0 | 0
Cardiac output decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac pacemaker evaluation (Investigations) | 1 | 1 | 0 | 0 | 1
Cardiac stress test (Investigations) | 2 | 1 | 2 | 0 | 1
Cardiac stress test abnormal (Investigations) | 3 | 1 | 1 | 1 | 0
Cardiovascular evaluation (Investigations) | 19 | 21 | 20 | 4 | 8
Cardiovascular function test (Investigations) | 0 | 0 | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Cholangiogram (Investigations) | 0 | 0 | 3 | 0 | 0
Coagulation test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Coagulation time prolonged (Investigations) | 2 | 0 | 0 | 0 | 0
Coagulation time shortened (Investigations) | 1 | 1 | 0 | 0 | 0
Colonoscopy (Investigations) | 18 | 14 | 6 | 3 | 6
Colonoscopy abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Colonoscopy normal (Investigations) | 1 | 0 | 0 | 0 | 0
Computerised tomogram (Investigations) | 2 | 0 | 0 | 0 | 0
Computerised tomogram abdomen (Investigations) | 1 | 1 | 0 | 0 | 0
Computerised tomogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Computerised tomogram thorax (Investigations) | 0 | 0 | 1 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Cyst aspiration (Investigations) | 1 | 0 | 0 | 0 | 0
Cystogram (Investigations) | 1 | 0 | 0 | 0 | 0
Cystoscopy (Investigations) | 4 | 13 | 12 | 1 | 2
Cystoscopy abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Dermatologic examination (Investigations) | 0 | 1 | 0 | 0 | 0
Diagnostic procedure (Investigations) | 1 | 7 | 10 | 2 | 3
Drug level decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Ear, nose and throat examination (Investigations) | 0 | 0 | 0 | 1 | 0
Echocardiogram (Investigations) | 1 | 1 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 1 | 1 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram ambulatory (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram change (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram normal (Investigations) | 1 | 1 | 0 | 0 | 0
Electroneuromyography (Investigations) | 0 | 0 | 1 | 0 | 0
Endocrine test (Investigations) | 0 | 0 | 1 | 0 | 0
Endoscopic retrograde cholangiopancreatography (Investigations) | 5 | 1 | 0 | 1 | 1
Endoscopy (Investigations) | 2 | 4 | 0 | 1 | 0
Endoscopy gastrointestinal (Investigations) | 0 | 1 | 1 | 0 | 0
Endoscopy upper gastrointestinal tract (Investigations) | 4 | 5 | 1 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 1 | 0 | 0 | 0
Flexible sigmoidoscopy (Investigations) | 1 | 0 | 1 | 0 | 0
Functional residual capacity decreased (Investigations) | 0 | 2 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Gynaecological examination (Investigations) | 0 | 0 | 0 | 1 | 0
HIV test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 4 | 1 | 0 | 1
Heart rate abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 1 | 2 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 2 | 0 | 0 | 0 | 0
Hysteroscopy (Investigations) | 0 | 1 | 0 | 1 | 1
International normalised ratio (Investigations) | 0 | 0 | 0 | 0 | 2
International normalised ratio decreased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 3 | 3 | 3 | 0 | 0
Investigation (Investigations) | 3 | 4 | 2 | 0 | 2
Laparoscopy (Investigations) | 1 | 0 | 2 | 0 | 0
Laryngoscopy (Investigations) | 1 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 2 | 1 | 2 | 0 | 1
Mean arterial pressure (Investigations) | 0 | 0 | 1 | 0 | 0
Mediastinoscopy (Investigations) | 0 | 1 | 3 | 0 | 0
Medical observation (Investigations) | 9 | 14 | 9 | 0 | 0
Medication residue (Investigations) | 0 | 0 | 0 | 1 | 0
Muscle relaxant drug level above therapeutic (Investigations) | 0 | 0 | 1 | 0 | 0
Neurological examination (Investigations) | 0 | 1 | 1 | 0 | 0
Nuclear magnetic resonance imaging (Investigations) | 2 | 0 | 2 | 0 | 0
Occult blood (Investigations) | 2 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 2 | 1 | 0 | 0
Oesophagogastroduodenoscopy (Investigations) | 2 | 2 | 2 | 1 | 2
Orthopedic examination (Investigations) | 0 | 1 | 0 | 0 | 0
Pain assessment (Investigations) | 1 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1 | 0 | 0
Platelet count increased (Investigations) | 1 | 1 | 0 | 0 | 0
Prostate examination (Investigations) | 0 | 1 | 0 | 0 | 0
Prothrombin level decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Prothrombin time shortened (Investigations) | 0 | 0 | 0 | 1 | 0
Psychiatric evaluation (Investigations) | 1 | 1 | 0 | 0 | 0
Pulmonary function challenge test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Pyelogram retrograde (Investigations) | 0 | 0 | 1 | 0 | 0
Pyelogram retrograde normal (Investigations) | 0 | 0 | 0 | 1 | 0
Sigmoidoscopy (Investigations) | 1 | 0 | 0 | 0 | 0
Sleep study (Investigations) | 2 | 3 | 3 | 0 | 2
Spinal X-ray (Investigations) | 0 | 1 | 0 | 0 | 0
Stress echocardiogram (Investigations) | 0 | 0 | 1 | 0 | 0
Transplant evaluation (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0
Ultrasound Doppler (Investigations) | 0 | 1 | 0 | 0 | 0
Ultrasound scan (Investigations) | 1 | 0 | 0 | 0 | 0
Ureteroscopy (Investigations) | 0 | 0 | 1 | 0 | 0
Urethroscopy (Investigations) | 0 | 0 | 1 | 0 | 0
Urodynamics measurement (Investigations) | 0 | 1 | 1 | 0 | 0
Urogram (Investigations) | 1 | 0 | 0 | 0 | 0
Urological examination (Investigations) | 0 | 1 | 0 | 0 | 0
Vascular test (Investigations) | 0 | 1 | 0 | 2 | 0
Weight decreased (Investigations) | 9 | 6 | 5 | 2 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
X-ray (Investigations) | 1 | 0 | 0 | 0 | 0
X-ray limb (Investigations) | 0 | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 8 | 3 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 57 | 32 | 37 | 6 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 304 | 394 | 361 | 195 | 239
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 2 | 2 | 1 | 3
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diet refusal (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 6 | 0 | 1 | 0
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 4 | 0 | 4 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 14 | 7 | 7 | 2 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 122 | 133 | 132 | 40 | 47
Hyperkalaemia (Metabolism and nutrition disorders) | 45 | 23 | 28 | 7 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperphagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 59 | 51 | 55 | 19 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 5 | 5 | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 21 | 8 | 20 | 6 | 5
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 4 | 2 | 3 | 0 | 0
Increased insulin requirement (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 9 | 6 | 7 | 1 | 4
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Lipomatosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 0
Marasmus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 4 | 2 | 1 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Neuroglycopenia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0
Podagra (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Salt intoxication (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 7 | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 10 | 5 | 2 | 2
Arthritis allergic (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 28 | 34 | 7 | 7
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 5 | 4 | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 1
Chondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 1 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 3 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 4 | 6 | 2 | 1 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 0 | 2
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 12 | 9 | 6 | 1 | 3
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1 | 0
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 7 | 11 | 1 | 4
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 2 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 15 | 13 | 9 | 2 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 8 | 9 | 3 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4 | 1 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Myopathy steroid (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 22 | 40 | 25 | 16 | 10
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 5 | 3 | 4 | 1 | 3
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 4 | 12 | 0 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 6 | 1 | 5 | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 2 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 5 | 4 | 5 | 1 | 1
Senile ankylosing vertebral hyperostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 | 9 | 7 | 2 | 4
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 | 9 | 10 | 8 | 4
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 2 | 0 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5 | 2 | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 2 | 0 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Anaplastic thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Angiocentric lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 58 | 53 | 52 | 7 | 9
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 1 | 2 | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36 | 47 | 38 | 12 | 13
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 7 | 1 | 3
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 4 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 10 | 21 | 2 | 4
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 | 30 | 36 | 19 | 16
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Carcinoma in situ of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Cerebral neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 5 | 0 | 0
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Chronic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 5 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 78 | 80 | 68 | 21 | 28
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cranial nerve neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Dysplastic naevus syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 1 | 1 | 0
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Epithelioid sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3 | 3 | 0 | 0
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 17 | 18 | 7 | 6
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Genitourinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0 | 0
Gum neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4 | 2 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 25 | 24 | 7 | 4
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Histiocytosis haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 8 | 8 | 3 | 2
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 8 | 8 | 1 | 3
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 0 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 2 | 0 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 110 | 102 | 109 | 30 | 23
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 14 | 14 | 6 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 19 | 17 | 2 | 4
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant mesenchymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 2 | 1 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant neoplasm of thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 3 | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5 | 6 | 0 | 2
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6 | 4 | 0 | 0
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Metastases to large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8 | 4 | 2 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7 | 3 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 2 | 0 | 0
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0 | 0
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 4 | 2 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7 | 2 | 3 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 3 | 0 | 3
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 1
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 3 | 1 | 1
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 7 | 8 | 1 | 0
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8 | 6 | 2 | 2
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 10 | 6 | 0 | 2
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Omentum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Oral cavity cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Oropharyngeal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 8 | 4 | 2
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 18 | 20 | 6 | 5
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 0 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Penile neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 1
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 | 0 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 132 | 136 | 119 | 34 | 24
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 3 | 1 | 1
Pseudomyxoma peritonei (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6 | 10 | 1 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Renal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 7 | 4
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 19 | 17 | 0 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 7 | 3 | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 92 | 100 | 102 | 22 | 19
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 12 | 15 | 3 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 3 | 1 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tendon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3 | 0 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 4 | 2 | 1
Tongue cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 2 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 3 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 1 | 0 | 1
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 2 | 0 | 0
Urethral cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 8 | 3 | 3 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 3
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 0 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 2 | 1 | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 3 | 1 | 0 | 0
Anaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anoxic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 2 | 3 | 0 | 1 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 2 | 1 | 1 | 0 | 0
Benign intracranial hypertension (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Brain mass (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Brain stem ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Carotid artery disease (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 4 | 1 | 4 | 1 | 1
Carotid sinus syndrome (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 2 | 6 | 0 | 1 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 2 | 1 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 2 | 0 | 2 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral circulatory failure (Nervous system disorders) | 0 | 0 | 2 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 32 | 34 | 44 | 8 | 16
Cerebral hypoperfusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 254 | 259 | 271 | 82 | 93
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 144 | 141 | 162 | 51 | 53
Cerebrovascular disorder (Nervous system disorders) | 1 | 2 | 0 | 1 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 2 | 0 | 2 | 0
Cervical root pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 2 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 15 | 15 | 9 | 6 | 5
Dementia (Nervous system disorders) | 16 | 6 | 16 | 4 | 1
Dementia Alzheimer's type (Nervous system disorders) | 6 | 2 | 2 | 0 | 2
Dementia of the Alzheimer's type, with delirium (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 4 | 1 | 3 | 1 | 0
Dizziness (Nervous system disorders) | 44 | 51 | 40 | 11 | 10
Dizziness exertional (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Drop attacks (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Encephalitis (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 5 | 6 | 9 | 1 | 5
Epilepsy (Nervous system disorders) | 6 | 8 | 10 | 5 | 3
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Facial palsy (Nervous system disorders) | 1 | 4 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 2 | 0 | 0 | 1 | 1
Global amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 1 | 3 | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 4 | 16 | 5 | 3 | 8
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 2 | 1 | 0 | 1 | 1
Hydrocephalus (Nervous system disorders) | 2 | 1 | 1 | 1 | 0
Hyperpathia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 2 | 2 | 1 | 1 | 4
Hypertonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Hypokinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 4 | 2 | 2 | 1 | 0
Hypotonic-hyporesponsive episode (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 2 | 0 | 2 | 0 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 3 | 0 | 0
Loss of consciousness (Nervous system disorders) | 4 | 6 | 3 | 1 | 2
Lumbar radiculopathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 2 | 2 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 2 | 1 | 1
Migraine (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Motor neurone disease (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myelitis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 2 | 1 | 0
Neuritis (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Neurodegenerative disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 4 | 3 | 3 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 2 | 2
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 1 | 2 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Paresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 5 | 6 | 0 | 1 | 1
Parkinsonism (Nervous system disorders) | 2 | 1 | 4 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Peripheral paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 3 | 0 | 3 | 2 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Post-traumatic epilepsy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Postictal state (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 16 | 14 | 13 | 2 | 4
Pseudobulbar palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Radicular pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Radicular syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Radiculitis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Radiculitis lumbosacral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 3 | 0 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 11 | 6 | 7 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Spinal cord ischaemia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Spinal epidural haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 6 | 10 | 7 | 0 | 2
Supranuclear palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 112 | 133 | 127 | 31 | 19
Syncope vasovagal (Nervous system disorders) | 14 | 13 | 13 | 2 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Tonic convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 192 | 183 | 199 | 57 | 60
Tremor (Nervous system disorders) | 0 | 2 | 2 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Vascular dementia (Nervous system disorders) | 1 | 1 | 3 | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 3 | 0 | 1 | 1
Vascular headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 3 | 6 | 3 | 1 | 5
Vertigo CNS origin (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Wernicke's encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Perineal haematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 9 | 5 | 4 | 4 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Cardiac neurosis (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Catatonia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 5 | 5 | 3 | 4 | 0
Conduct disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 14 | 11 | 5 | 3 | 4
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 4 | 1 | 3 | 1 | 1
Delirium tremens (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Delusional disorder, persecutory type (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 20 | 20 | 13 | 4 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Emotional distress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 1 | 3 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 2 | 2 | 0 | 0 | 2
Mental disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 7 | 9 | 8 | 2 | 3
Narcissistic personality disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Neurosis (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 3 | 0 | 1 | 0 | 0
Personality change due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Phobia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Psychosomatic disease (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 3 | 0 | 2 | 1 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 6 | 6 | 2 | 0 | 1
Anuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 3 | 4 | 0 | 0 | 2
Bladder cyst (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0
Bladder dilatation (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bladder mass (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Bladder neck sclerosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 2 | 1 | 2 | 0 | 0
Bladder stenosis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 4 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 4 | 3 | 1 | 0 | 1
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 7 | 5 | 6 | 3 | 3
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0
Diabetic end stage renal disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 192 | 181 | 180 | 57 | 61
Dysuria (Renal and urinary disorders) | 1 | 6 | 2 | 0 | 0
Enuresis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Glomerulonephritis proliferative (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Glomerulosclerosis (Renal and urinary disorders) | 3 | 4 | 5 | 2 | 0
Haematuria (Renal and urinary disorders) | 19 | 18 | 24 | 3 | 4
Hydronephrosis (Renal and urinary disorders) | 2 | 3 | 3 | 2 | 1
Hypertensive nephropathy (Renal and urinary disorders) | 15 | 8 | 14 | 8 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Kidney fibrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 1 | 2 | 3 | 0 | 0
Nephritis (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0
Nephritis interstitial (Renal and urinary disorders) | 1 | 1 | 1 | 2 | 1
Nephroangiosclerosis (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 19 | 18 | 22 | 7 | 4
Nephropathy (Renal and urinary disorders) | 4 | 3 | 5 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 3 | 6 | 2 | 1 | 2
Nephrosclerosis (Renal and urinary disorders) | 6 | 3 | 5 | 5 | 1
Nephrotic syndrome (Renal and urinary disorders) | 2 | 5 | 1 | 0 | 2
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 3 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 5 | 2 | 2
Renal aneurysm (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0
Renal artery arteriosclerosis (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0
Renal artery occlusion (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 9 | 6 | 3 | 1 | 6
Renal atrophy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 5 | 4 | 5 | 3 | 1
Renal cyst (Renal and urinary disorders) | 4 | 2 | 1 | 0 | 2
Renal disorder (Renal and urinary disorders) | 3 | 1 | 2 | 0 | 0
Renal embolism (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 140 | 115 | 107 | 23 | 19
Renal failure acute (Renal and urinary disorders) | 61 | 36 | 29 | 7 | 11
Renal failure chronic (Renal and urinary disorders) | 25 | 11 | 10 | 5 | 6
Renal impairment (Renal and urinary disorders) | 20 | 18 | 13 | 8 | 3
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal ischaemia (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Renal mass (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Renal tubular acidosis (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0
Renal vessel disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Residual urine (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urate nephropathy (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Ureteral disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 0
Urethral dilatation (Renal and urinary disorders) | 1 | 3 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 5 | 4 | 2 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 2 | 1 | 1
Urinary retention (Renal and urinary disorders) | 12 | 17 | 25 | 3 | 4
Urinary tract disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract inflammation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 3 | 0 | 3 | 1 | 0
Urinoma (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Vesical fistula (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 25 | 30 | 25 | 3 | 6
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Breast dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Breast inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Calculus prostatic (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 1 | 2 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0 | 1 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Genital prolapse (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 2 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Orchitis noninfective (Reproductive system and breast disorders) | 1 | 0 | 4 | 0 | 0
Organic erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2 | 1 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Peyronie's disease (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Prostatic atrophy (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Prostatic disorder (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0 | 3 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 3 | 6 | 1 | 4 | 1
Prostatomegaly (Reproductive system and breast disorders) | 5 | 2 | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Testicular mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Urogenital prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine cervical erosion (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Uterine cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Uterine disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Uterine fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 2 | 0 | 0 | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Vaginal lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vulval ulceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 12 | 2 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 5 | 1 | 2
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Alveolitis fibrosing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Anoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 23 | 17 | 22 | 11 | 12
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchial polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 7 | 8 | 7
Broncholithiasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchopulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 52 | 61 | 66 | 16 | 24
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 6 | 11 | 1 | 4
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 50 | 51 | 52 | 12 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 10 | 12 | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 8 | 3 | 7
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 4 | 1 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 2 | 0
Laryngitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 7 | 3 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 19 | 3 | 3
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 6 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 4 | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4 | 3 | 0
Pneumothorax spontaneous tension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 41 | 50 | 35 | 14 | 14
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 8 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 12 | 6 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 23 | 24 | 33 | 5 | 7
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 10 | 14 | 15 | 1 | 8
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Wegener's granulomatosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 8 | 5 | 16 | 1 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Cutaneous amyloidosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 2 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 108 | 121 | 114 | 18 | 19
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Parapsoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 2 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 285 | 314 | 321 | 74 | 59
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0 | 1
Alcohol use (Social circumstances) | 0 | 1 | 1 | 0 | 0
Cardiac assistance device user (Social circumstances) | 0 | 0 | 1 | 0 | 0
Cardiac valve prosthesis user (Social circumstances) | 1 | 0 | 0 | 0 | 0
Death of relative (Social circumstances) | 0 | 0 | 1 | 0 | 0
Exercise adequate (Social circumstances) | 0 | 1 | 0 | 0 | 0
Hearing disability (Social circumstances) | 0 | 0 | 0 | 1 | 0
Homicide (Social circumstances) | 1 | 1 | 0 | 0 | 0
Joint prosthesis user (Social circumstances) | 1 | 1 | 1 | 0 | 0
Limb prosthesis user (Social circumstances) | 1 | 1 | 0 | 0 | 0
Living in residential institution (Social circumstances) | 0 | 1 | 0 | 0 | 0
Overwork (Social circumstances) | 1 | 0 | 0 | 0 | 0
Physical assault (Social circumstances) | 1 | 0 | 0 | 0 | 0
Refusal of treatment by patient (Social circumstances) | 0 | 1 | 1 | 1 | 0
Respite care (Social circumstances) | 1 | 0 | 0 | 0 | 0
Sexual relationship change (Social circumstances) | 0 | 1 | 0 | 0 | 0
Social stay hospitalisation (Social circumstances) | 9 | 6 | 3 | 1 | 4
Treatment noncompliance (Social circumstances) | 2 | 2 | 2 | 3 | 1
Victim of crime (Social circumstances) | 0 | 0 | 1 | 0 | 0
Walking disability (Social circumstances) | 1 | 0 | 0 | 0 | 0
Abdominal cavity drainage (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Abdominal hernia repair (Surgical and medical procedures) | 4 | 5 | 2 | 0 | 1
Abdominal operation (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 1
Abdominoplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Abscess drainage (Surgical and medical procedures) | 1 | 3 | 4 | 1 | 0
Adenoidectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Adhesiolysis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Alcohol rehabilitation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Amputation (Surgical and medical procedures) | 34 | 47 | 39 | 6 | 6
Amputation of penis (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Amputation revision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Anal fissure excision (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
Anal fistula excision (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Anal lesion excision (Surgical and medical procedures) | 1 | 1 | 2 | 0 | 1
Anal sphincterotomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Analgesic intervention supportive therapy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Analgesic therapy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Angioplasty (Surgical and medical procedures) | 346 | 333 | 317 | 71 | 68
Ankle arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Ankle operation (Surgical and medical procedures) | 0 | 1 | 2 | 0 | 1
Ankle reconstruction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Antibiotic prophylaxis (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Anticoagulant therapy (Surgical and medical procedures) | 3 | 1 | 1 | 0 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 18 | 17 | 14 | 1 | 1
Aortic bypass (Surgical and medical procedures) | 4 | 3 | 3 | 0 | 1
Aortic surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 2
Aortic valve repair (Surgical and medical procedures) | 4 | 2 | 7 | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 17 | 30 | 24 | 6 | 13
Appendicectomy (Surgical and medical procedures) | 6 | 5 | 11 | 1 | 2
Arterial aneurysm repair (Surgical and medical procedures) | 1 | 1 | 1 | 0 | 1
Arterial bypass operation (Surgical and medical procedures) | 6 | 3 | 4 | 0 | 1
Arterial stent insertion (Surgical and medical procedures) | 3 | 2 | 5 | 1 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0
Arteriovenous graft (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Arteriovenous shunt operation (Surgical and medical procedures) | 1 | 0 | 3 | 0 | 0
Arthrodesis (Surgical and medical procedures) | 0 | 4 | 1 | 0 | 1
Arthroscopic surgery (Surgical and medical procedures) | 1 | 2 | 1 | 0 | 0
Artificial urinary sphincter implant (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Atrial septal defect repair (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Balneotherapy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Benign tumour excision (Surgical and medical procedures) | 2 | 0 | 0 | 1 | 0
Bilateral orchidectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Bile duct T-tube removal (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Biliary tract operation (Surgical and medical procedures) | 3 | 0 | 1 | 0 | 0
Bladder catheterisation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Bladder lesion excision (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Bladder neck resection (Surgical and medical procedures) | 1 | 2 | 0 | 0 | 0
Bladder neoplasm surgery (Surgical and medical procedures) | 1 | 2 | 2 | 1 | 0
Bladder operation (Surgical and medical procedures) | 1 | 4 | 1 | 0 | 0
Bladder polypectomy (Surgical and medical procedures) | 0 | 3 | 1 | 0 | 0
Bladder repair (Surgical and medical procedures) | 1 | 4 | 1 | 1 | 0
Bladder sphincterectomy (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Blood pressure management (Surgical and medical procedures) | 1 | 1 | 1 | 0 | 1
Bone debridement (Surgical and medical procedures) | 1 | 1 | 1 | 0 | 0
Bone operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Brachytherapy (Surgical and medical procedures) | 2 | 1 | 1 | 0 | 1
Brachytherapy to prostate (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Brachytherapy to uterus (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Brain operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Breast operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Bunion operation (Surgical and medical procedures) | 3 | 4 | 3 | 1 | 3
Burn debridement (Surgical and medical procedures) | 0 | 0 | 2 | 0 | 0
Bursa removal (Surgical and medical procedures) | 0 | 2 | 1 | 0 | 0
Cardiac ablation (Surgical and medical procedures) | 2 | 7 | 2 | 1 | 1
Cardiac aneurysm repair (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 4 | 6 | 4 | 0 | 2
Cardiac pacemaker insertion (Surgical and medical procedures) | 56 | 62 | 69 | 13 | 20
Cardiac pacemaker removal (Surgical and medical procedures) | 1 | 1 | 3 | 0 | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 10 | 9 | 8 | 2 | 4
Cardiac pacemaker revision (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 1
Cardiac rehabilitation therapy (Surgical and medical procedures) | 10 | 14 | 14 | 3 | 1
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 | 0 | 1 | 1 | 0
Cardiovascular event prophylaxis (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 4
Cardioversion (Surgical and medical procedures) | 2 | 4 | 0 | 1 | 1
Carotid endarterectomy (Surgical and medical procedures) | 72 | 84 | 62 | 16 | 16
Carpal tunnel decompression (Surgical and medical procedures) | 2 | 5 | 3 | 0 | 2
Cataract operation (Surgical and medical procedures) | 522 | 565 | 575 | 145 | 158
Catheter removal (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Catheterisation cardiac (Surgical and medical procedures) | 23 | 22 | 20 | 7 | 4
Cerebral decompression (Surgical and medical procedures) | 1 | 1 | 0 | 1 | 0
Cervical polypectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Cervix operation (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
Chemotherapy (Surgical and medical procedures) | 7 | 10 | 5 | 0 | 1
Chest tube insertion (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 49 | 62 | 80 | 22 | 17
Cholecystostomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Choledocholithotomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Choledochostomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Choledochotomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Cholelithotomy (Surgical and medical procedures) | 0 | 1 | 5 | 1 | 1
Chondroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Circumcision (Surgical and medical procedures) | 0 | 0 | 2 | 1 | 0
Colectomy (Surgical and medical procedures) | 6 | 11 | 8 | 1 | 2
Colectomy total (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Colon operation (Surgical and medical procedures) | 0 | 3 | 0 | 1 | 0
Colon polypectomy (Surgical and medical procedures) | 4 | 1 | 1 | 1 | 2
Colostomy (Surgical and medical procedures) | 4 | 5 | 3 | 0 | 1
Colostomy closure (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Colporrhaphy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Colposuspension (Surgical and medical procedures) | 1 | 1 | 0 | 1 | 0
Corneal operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Corneal transplant (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 606 | 645 | 617 | 198 | 211
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 2 | 3 | 0 | 0
Coronary artery bypass (Surgical and medical procedures) | 240 | 260 | 271 | 79 | 83
Coronary revascularisation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Cox-Maze procedure (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Cranial nerve operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Craniotomy (Surgical and medical procedures) | 0 | 2 | 0 | 0 | 0
Cyst drainage (Surgical and medical procedures) | 0 | 0 | 2 | 0 | 0
Cyst removal (Surgical and medical procedures) | 0 | 2 | 5 | 1 | 0
Cystocele repair (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 1
Cystopexy (Surgical and medical procedures) | 1 | 0 | 1 | 1 | 1
Cystoprostatectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Cystostomy (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0
Dacryocystorhinostomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Debridement (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Dental implantation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Dental operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Detoxification (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus management (Surgical and medical procedures) | 9 | 12 | 8 | 6 | 7
Dialysis (Surgical and medical procedures) | 42 | 31 | 29 | 6 | 8
Diathermy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Drug therapy (Surgical and medical procedures) | 1 | 2 | 4 | 1 | 2
Drug therapy changed (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Duodenal sphincterotomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Duodenectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Dupuytren's contracture operation (Surgical and medical procedures) | 3 | 4 | 2 | 0 | 2
Ear operation (Surgical and medical procedures) | 4 | 1 | 0 | 1 | 0
Elective surgery (Surgical and medical procedures) | 0 | 0 | 2 | 0 | 0
Electron radiation therapy to prostate (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Empyema drainage (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Endarterectomy (Surgical and medical procedures) | 5 | 2 | 3 | 0 | 1
Endarterectomy of aorta (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Endometrial ablation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Epididymal cyst removal (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Epididymal operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Ethmoid sinus surgery (Surgical and medical procedures) | 2 | 0 | 2 | 0 | 0
Eventration procedure (Surgical and medical procedures) | 1 | 4 | 1 | 1 | 0
Excision of palatal lesion (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Explorative laparotomy (Surgical and medical procedures) | 0 | 2 | 0 | 0 | 0
Exploratory operation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Eye laser surgery (Surgical and medical procedures) | 2 | 1 | 0 | 0 | 1
Eye operation (Surgical and medical procedures) | 2 | 8 | 3 | 2 | 3
Eyelid operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Face lift (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1
Fasciectomy (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Fasciotomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Femoral hernia repair (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Finger amputation (Surgical and medical procedures) | 2 | 1 | 2 | 0 | 1
Fistula repair (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 1
Fluid intake restriction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Foot amputation (Surgical and medical procedures) | 1 | 4 | 1 | 0 | 0
Foot operation (Surgical and medical procedures) | 1 | 2 | 5 | 0 | 0
Fracture debridement (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Fracture reduction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Frontal sinus operation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Gallbladder operation (Surgical and medical procedures) | 2 | 2 | 9 | 1 | 0
Gastrectomy (Surgical and medical procedures) | 0 | 3 | 1 | 0 | 2
Gastric banding (Surgical and medical procedures) | 1 | 2 | 0 | 0 | 1
Gastric bypass (Surgical and medical procedures) | 1 | 2 | 1 | 0 | 0
Gastric operation (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
Gastric polypectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Gastro-jejunostomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Gastrointestinal tube insertion (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Gastrostomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Gastrostomy tube insertion (Surgical and medical procedures) | 1 | 1 | 0 | 1 | 0
General anaesthesia (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Genitourinary operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1
Gingival operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Glaucoma surgery (Surgical and medical procedures) | 0 | 2 | 3 | 0 | 1
Haematoma evacuation (Surgical and medical procedures) | 2 | 1 | 0 | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 8 | 5 | 8 | 2 | 5
Heart valve operation (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Heel nodule excision (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Heparin neutralisation therapy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Hepatectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1
Hepaticojejunostomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Hernia hiatus repair (Surgical and medical procedures) | 0 | 1 | 2 | 1 | 1
Hernia repair (Surgical and medical procedures) | 23 | 27 | 23 | 2 | 6
High frequency ablation (Surgical and medical procedures) | 1 | 1 | 4 | 2 | 4
Hip arthroplasty (Surgical and medical procedures) | 59 | 91 | 62 | 17 | 21
Hip surgery (Surgical and medical procedures) | 7 | 8 | 11 | 3 | 3
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 0 | 2 | 2
Hydrocele excision (Surgical and medical procedures) | 0 | 7 | 0 | 0 | 0
Hydrocele repair (Surgical and medical procedures) | 0 | 1 | 2 | 0 | 1
Hypotensive anaesthesia procedure (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 9 | 8 | 5 | 4 | 4
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Ileectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Ileostomy (Surgical and medical procedures) | 1 | 2 | 1 | 0 | 0
Ileostomy closure (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 13 | 25 | 12 | 1 | 3
Implantable defibrillator replacement (Surgical and medical procedures) | 4 | 1 | 2 | 0 | 0
Incisional drainage (Surgical and medical procedures) | 0 | 0 | 2 | 0 | 0
Incisional hernia repair (Surgical and medical procedures) | 2 | 6 | 5 | 1 | 1
Indwelling catheter management (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 48 | 54 | 40 | 14 | 15
Internal fixation of fracture (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Intervertebral disc operation (Surgical and medical procedures) | 14 | 10 | 11 | 1 | 3
Intestinal adhesion lysis (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Intestinal anastomosis (Surgical and medical procedures) | 0 | 2 | 0 | 1 | 1
Intestinal fistula repair (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Intestinal operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Intestinal polypectomy (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Intestinal resection (Surgical and medical procedures) | 1 | 2 | 0 | 0 | 1
Intestinal stent insertion (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Intestinal stoma (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Intraocular lens extraction (Surgical and medical procedures) | 1 | 4 | 0 | 0 | 1
Intraocular lens implant (Surgical and medical procedures) | 0 | 2 | 4 | 0 | 2
Isotope therapy to thyroid (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Joint arthroplasty (Surgical and medical procedures) | 5 | 4 | 4 | 2 | 0
Joint injection (Surgical and medical procedures) | 1 | 0 | 1 | 1 | 0
Joint irrigation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Joint manipulation (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Joint reconstruction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Joint resurfacing surgery (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Joint surgery (Surgical and medical procedures) | 1 | 2 | 2 | 0 | 0
Keratoplasty (Surgical and medical procedures) | 0 | 0 | 1 | 1 | 0
Kidney anastomosis (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 73 | 97 | 80 | 28 | 30
Knee meniscectomy (Surgical and medical procedures) | 1 | 1 | 0 | 2 | 1
Knee operation (Surgical and medical procedures) | 11 | 13 | 12 | 5 | 4
Laparoscopic surgery (Surgical and medical procedures) | 3 | 1 | 1 | 0 | 0
Laparotomy (Surgical and medical procedures) | 2 | 2 | 0 | 0 | 0
Large intestine anastomosis (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Laryngeal operation (Surgical and medical procedures) | 1 | 1 | 1 | 0 | 0
Laryngectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Laser therapy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Leg amputation (Surgical and medical procedures) | 5 | 7 | 1 | 0 | 0
Lesion excision (Surgical and medical procedures) | 2 | 0 | 2 | 0 | 0
Ligament operation (Surgical and medical procedures) | 0 | 1 | 1 | 1 | 0
Limb operation (Surgical and medical procedures) | 2 | 3 | 2 | 0 | 1
Lip lesion excision (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Lip operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Lipoma excision (Surgical and medical procedures) | 2 | 1 | 2 | 2 | 0
Liposuction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Liver operation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Lung cyst removal (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Lung lobectomy (Surgical and medical procedures) | 1 | 2 | 2 | 0 | 0
Lung operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Lymphadenectomy (Surgical and medical procedures) | 2 | 0 | 1 | 1 | 0
Malignant tumour excision (Surgical and medical procedures) | 0 | 3 | 0 | 0 | 1
Mandibulectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Mass excision (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Mastectomy (Surgical and medical procedures) | 2 | 4 | 1 | 1 | 0
Maxillary antrum operation (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Mediastinal operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Medical device implantation (Surgical and medical procedures) | 0 | 0 | 2 | 0 | 1
Medical device removal (Surgical and medical procedures) | 4 | 2 | 3 | 1 | 2
Medical diet (Surgical and medical procedures) | 2 | 1 | 0 | 0 | 0
Meningioma surgery (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Meniscus operation (Surgical and medical procedures) | 1 | 2 | 6 | 0 | 2
Mitral valve repair (Surgical and medical procedures) | 4 | 0 | 7 | 0 | 2
Mitral valve replacement (Surgical and medical procedures) | 7 | 5 | 8 | 3 | 1
Modified radical mastectomy (Surgical and medical procedures) | 0 | 0 | 2 | 0 | 0
Myringoplasty (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 1
Nail operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Nasal cyst removal (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Nasal operation (Surgical and medical procedures) | 1 | 4 | 2 | 0 | 2
Nasal polypectomy (Surgical and medical procedures) | 2 | 2 | 1 | 1 | 0
Nasal septal operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Neck exploration (Surgical and medical procedures) | 1 | 0 | 1 | 1 | 0
Nephrectomy (Surgical and medical procedures) | 3 | 3 | 2 | 2 | 0
Nephrostomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Nephroureterectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Nerve block (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Nervous system surgery (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Neurectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Neurolysis (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Oesophageal dilation procedure (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Oesophageal operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Oesophagogastric fundoplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Oophorectomy bilateral (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1
Open reduction of fracture (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Orchidectomy (Surgical and medical procedures) | 0 | 2 | 0 | 0 | 1
Orthopedic procedure (Surgical and medical procedures) | 6 | 1 | 7 | 0 | 2
Ossicular operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Ostectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Osteomyelitis drainage (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Osteosynthesis (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Osteotomy (Surgical and medical procedures) | 2 | 1 | 0 | 1 | 0
Otorhinolaryngological surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Ovarian operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Packed red blood cell transfusion (Surgical and medical procedures) | 0 | 3 | 0 | 0 | 0
Pain management (Surgical and medical procedures) | 1 | 3 | 0 | 0 | 0
Palliative care (Surgical and medical procedures) | 2 | 2 | 2 | 0 | 1
Pancreatic operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Pancreaticoduodenectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Pancreaticosplenectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Papilloma excision (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Parathyroid gland operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Parathyroidectomy (Surgical and medical procedures) | 4 | 3 | 2 | 0 | 1
Parotidectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Pelvic exploration (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Penile prosthesis insertion (Surgical and medical procedures) | 1 | 2 | 3 | 0 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 3 | 0 | 1 | 0 | 1
Perineoplasty (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0
Peripheral artery angioplasty (Surgical and medical procedures) | 2 | 2 | 0 | 0 | 0
Peripheral nerve decompression (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Peripheral nerve operation (Surgical and medical procedures) | 1 | 1 | 1 | 0 | 0
Peripheral revascularisation (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Peritoneal dialysis (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
Peritoneal lavage (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Phlebectomy (Surgical and medical procedures) | 1 | 2 | 2 | 2 | 3
Physiotherapy (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Pilonidal sinus repair (Surgical and medical procedures) | 0 | 1 | 0 | 1 | 0
Plastic surgery (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 1
Polypectomy (Surgical and medical procedures) | 2 | 2 | 3 | 1 | 0
Postoperative analgesia (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Postoperative care (Surgical and medical procedures) | 0 | 1 | 4 | 1 | 0
Preoperative care (Surgical and medical procedures) | 0 | 4 | 2 | 0 | 0
Prolapse repair (Surgical and medical procedures) | 0 | 1 | 1 | 1 | 0
Prophylaxis (Surgical and medical procedures) | 9 | 10 | 7 | 2 | 0
Prophylaxis against gastrointestinal ulcer (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Prophylaxis of nausea and vomiting (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Prostatectomy (Surgical and medical procedures) | 20 | 23 | 21 | 9 | 5
Prostatic operation (Surgical and medical procedures) | 2 | 0 | 1 | 0 | 1
Prosthesis implantation (Surgical and medical procedures) | 2 | 2 | 3 | 0 | 0
Pyelolithotomy (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0
Radical mastectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Radical prostatectomy (Surgical and medical procedures) | 1 | 3 | 5 | 0 | 0
Radiculotomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Radioactive iodine therapy (Surgical and medical procedures) | 1 | 0 | 3 | 0 | 0
Radiotherapy (Surgical and medical procedures) | 0 | 2 | 3 | 1 | 0
Radiotherapy to liver (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Radiotherapy to prostate (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Rectal lesion excision (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Rectal polypectomy (Surgical and medical procedures) | 1 | 3 | 1 | 0 | 0
Rectal prolapse repair (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Rectocele repair (Surgical and medical procedures) | 0 | 4 | 0 | 1 | 0
Rehabilitation therapy (Surgical and medical procedures) | 27 | 22 | 34 | 9 | 9
Removal of foreign body (Surgical and medical procedures) | 1 | 1 | 1 | 1 | 0
Removal of foreign body from throat (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Removal of internal fixation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Renal artery stent placement (Surgical and medical procedures) | 2 | 0 | 2 | 0 | 0
Renal cyst excision (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Renal stone removal (Surgical and medical procedures) | 2 | 4 | 2 | 1 | 0
Renal surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Renal tumour excision (Surgical and medical procedures) | 1 | 0 | 1 | 1 | 0
Resection of rectum (Surgical and medical procedures) | 3 | 0 | 0 | 0 | 0
Resuscitation (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0
Retinal laser coagulation (Surgical and medical procedures) | 181 | 189 | 201 | 39 | 36
Retinal operation (Surgical and medical procedures) | 4 | 3 | 0 | 1 | 0
Revision of internal fixation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Rhinoplasty (Surgical and medical procedures) | 1 | 1 | 3 | 0 | 0
Rib excision (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Rotator cuff repair (Surgical and medical procedures) | 5 | 7 | 13 | 2 | 1
Routine health maintenance (Surgical and medical procedures) | 1 | 4 | 2 | 1 | 1
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Sebaceous cyst excision (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Septoplasty (Surgical and medical procedures) | 2 | 0 | 2 | 1 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 4 | 8 | 9 | 0 | 1
Shoulder operation (Surgical and medical procedures) | 3 | 7 | 5 | 2 | 3
Sigmoidectomy (Surgical and medical procedures) | 3 | 0 | 3 | 1 | 0
Sinus operation (Surgical and medical procedures) | 3 | 0 | 2 | 0 | 0
Skin cyst excision (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Skin graft (Surgical and medical procedures) | 0 | 0 | 4 | 0 | 0
Skin implant (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Skin lesion excision (Surgical and medical procedures) | 0 | 3 | 0 | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1 | 3 | 0 | 0
Small intestinal resection (Surgical and medical procedures) | 2 | 1 | 2 | 0 | 0
Speech rehabilitation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Sphenoid sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Spinal cord operation (Surgical and medical procedures) | 1 | 0 | 5 | 1 | 0
Spinal decompression (Surgical and medical procedures) | 6 | 9 | 5 | 0 | 2
Spinal deformity correction (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 5 | 4 | 8 | 3 | 2
Spinal laminectomy (Surgical and medical procedures) | 16 | 12 | 16 | 3 | 10
Spinal operation (Surgical and medical procedures) | 3 | 2 | 5 | 1 | 0
Spinal rod removal (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Splenectomy (Surgical and medical procedures) | 1 | 2 | 1 | 0 | 0
Stapedectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Stem cell transplant (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Stent placement (Surgical and medical procedures) | 9 | 7 | 4 | 2 | 1
Sternal wiring (Surgical and medical procedures) | 0 | 2 | 0 | 0 | 0
Steroid therapy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Strangulated hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Subdural haematoma evacuation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Suprapubic catheter insertion (Surgical and medical procedures) | 2 | 0 | 2 | 0 | 0
Surgery (Surgical and medical procedures) | 10 | 8 | 7 | 1 | 2
Suture removal (Surgical and medical procedures) | 1 | 2 | 0 | 1 | 0
Sympathectomy (Surgical and medical procedures) | 8 | 3 | 2 | 0 | 0
Synovectomy (Surgical and medical procedures) | 0 | 1 | 2 | 0 | 1
Tendon operation (Surgical and medical procedures) | 4 | 2 | 0 | 0 | 0
Tendon sheath lesion excision (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Tenotomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Testicular operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Therapeutic embolisation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Therapeutic procedure (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Therapy cessation (Surgical and medical procedures) | 2 | 9 | 1 | 1 | 0
Therapy regimen changed (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1
Thoracic cavity drainage (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Thoracotomy (Surgical and medical procedures) | 3 | 1 | 1 | 0 | 0
Thrombectomy (Surgical and medical procedures) | 2 | 2 | 1 | 0 | 0
Thromboembolectomy (Surgical and medical procedures) | 1 | 1 | 3 | 0 | 0
Thrombolysis (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Thyroglossal cyst excision (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Thyroid operation (Surgical and medical procedures) | 1 | 2 | 0 | 0 | 0
Thyroidectomy (Surgical and medical procedures) | 6 | 8 | 8 | 6 | 2
Toe amputation (Surgical and medical procedures) | 7 | 14 | 7 | 3 | 0
Toe operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 2 | 2 | 3 | 0 | 0
Trabeculectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Tracheal fistula repair (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Transfusion (Surgical and medical procedures) | 4 | 1 | 4 | 1 | 0
Transurethral bladder resection (Surgical and medical procedures) | 1 | 3 | 2 | 0 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 47 | 55 | 52 | 10 | 8
Tricuspid valve repair (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Tubal ligation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Tumour excision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Turbinectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Umbilical hernia repair (Surgical and medical procedures) | 5 | 10 | 4 | 0 | 1
Ureteral stent insertion (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Ureterectomy (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Ureteric calculus removal (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Ureterocelectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Ureterolithotomy (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Urethral dilation procedure (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Urethral operation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Urethral repair (Surgical and medical procedures) | 1 | 1 | 1 | 0 | 0
Urethral stent insertion (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Urethrotomy (Surgical and medical procedures) | 2 | 1 | 3 | 0 | 2
Urinary bladder excision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Urogenital fistula repair (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Uterine dilation and curettage (Surgical and medical procedures) | 2 | 2 | 1 | 1 | 2
Uterine prolapse repair (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Vaginal operation (Surgical and medical procedures) | 2 | 1 | 2 | 0 | 0
Vaginoperineorrhaphy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Vaginoplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1
Varicocele repair (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Varicose vein operation (Surgical and medical procedures) | 4 | 2 | 5 | 2 | 1
Vascular graft (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Vasectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Vasodilation procedure (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0
Venous ligation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 1
Venous operation (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Ventricular assist device insertion (Surgical and medical procedures) | 0 | 2 | 0 | 0 | 0
Vertebroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 2 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 5 | 4 | 3 | 1
Wedge resection toenail (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Weight loss diet (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Wound debridement (Surgical and medical procedures) | 3 | 1 | 1 | 0 | 0
Wrist surgery (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Accelerated hypertension (Vascular disorders) | 0 | 3 | 5 | 1 | 2
Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Aneurysm ruptured (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Angiopathy (Vascular disorders) | 1 | 4 | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 18 | 23 | 20 | 6 | 5
Aortic aneurysm rupture (Vascular disorders) | 5 | 8 | 9 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 2 | 2 | 0 | 0
Aortic dilatation (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 1 | 3 | 3 | 0
Aortic embolus (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aortic necrosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 3 | 2 | 2 | 1 | 2
Aortic thrombosis (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Arterial disorder (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 0 | 2 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 3 | 3 | 2 | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 2 | 0 | 0 | 0
Arterial stenosis limb (Vascular disorders) | 1 | 1 | 0 | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 2 | 2 | 0
Arteriosclerosis (Vascular disorders) | 5 | 8 | 11 | 4 | 2
Arteriosclerosis obliterans (Vascular disorders) | 1 | 4 | 2 | 0 | 0
Arteritis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 1 | 2 | 0 | 0 | 0
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Cardiovascular insufficiency (Vascular disorders) | 1 | 1 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 5 | 5 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 22 | 27 | 25 | 4 | 3
Diabetic macroangiopathy (Vascular disorders) | 0 | 2 | 1 | 0 | 0
Diabetic microangiopathy (Vascular disorders) | 0 | 3 | 0 | 0 | 0
Embolism (Vascular disorders) | 7 | 1 | 8 | 1 | 2
Essential hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1 | 2 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 1 | 2 | 1 | 0
Haematoma (Vascular disorders) | 2 | 5 | 1 | 5 | 1
Haemodynamic instability (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 11 | 7 | 4 | 5 | 3
Hypertension (Vascular disorders) | 97 | 84 | 94 | 33 | 42
Hypertensive crisis (Vascular disorders) | 8 | 8 | 17 | 4 | 8
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 83 | 57 | 55 | 15 | 13
Hypovolaemic shock (Vascular disorders) | 1 | 6 | 1 | 1 | 1
Iliac artery embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 689 | 686 | 657 | 198 | 168
Ischaemia (Vascular disorders) | 5 | 4 | 7 | 0 | 1
Ischaemic limb pain (Vascular disorders) | 1 | 1 | 1 | 0 | 0
Labile blood pressure (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Leriche syndrome (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Lymphostasis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Malignant hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 0
Microangiopathy (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Necrosis ischaemic (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Neurogenic shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 19 | 13 | 16 | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 9 | 5 | 7 | 2 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 2 | 3 | 0 | 0
Peripheral embolism (Vascular disorders) | 2 | 2 | 1 | 3 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 3 | 5 | 2 | 3
Peripheral vascular disorder (Vascular disorders) | 2 | 2 | 4 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 3 | 1 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Secondary hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 3 | 1 | 3 | 2 | 2
Shock haemorrhagic (Vascular disorders) | 2 | 1 | 1 | 0 | 0
Subclavian steal syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 0 | 1 | 2 | 0 | 0
Thrombophlebitis (Vascular disorders) | 4 | 3 | 7 | 2 | 2
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 5 | 1 | 2 | 1 | 0
Varicose ulceration (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 2 | 0 | 4
Vascular pseudoaneurysm (Vascular disorders) | 0 | 1 | 3 | 0 | 0
Vascular shunt (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Vascular stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Vasculitis necrotising (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Vasodilatation (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Venous stasis (Vascular disorders) | 1 | 1 | 1 | 1 | 2
Venous thrombosis (Vascular disorders) | 4 | 1 | 5 | 2 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 2 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
Only non-serious Adverse Events (AE) which lead to discontinuation of study medication were assessed and collected; the frequency was under 5%. Non-serious AEs per se were not assessed or collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.